**Study ID:** 213749

**Official Title of Study:** A Phase 1/2 randomized, observer-blinded, multi-country study to evaluate safety and immunogenicity of investigational adjuvanted human papillomavirus vaccine in females (16 to 26 years of age)

NCT number: NCT05496231

**Date of Document:** 08 FEB 2024


## STATISTICAL ANALYSIS PLAN

# 213749 (HPV9-AS04-001)

A Phase 1/2 randomized, observer-blinded, multi-country study to evaluate safety and immunogenicity of investigational adjuvanted human papillomavirus vaccine in females (16 to 26 years of age)

AUTHOR: PPD

VERSION NUMBER AND DATE: V3.0, 02FEB2024

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 Document:

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx

Author: PPD Version Number: 3.0

> Version Date: 02FEB2024

Template No.: CS\_TP\_BS016 Revision 7 Reference: CS WI BS005


## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V3.0 (Dated 02FEB2024) for Protocol 213749 (HPV9-AS04-001)

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|-------|-----------|------------------|
| Author: | PPD | Refe PPD | ebruary 6, 2024 |
| Position: | PPD | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|--------------|------------------------|-----------|------------------|
| Approved By: | PPD | PPD | Jary 8, 2024 |
| Position: | Senior Biostatistician | | |
| Company: | IQVIA | | |
| Approved By: | PPD | PPD | bruary 5, 2024 |
| Position: | Project Statistician | | |
| Company: | GSK | | |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the Document Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| 1.0 | 25APR2022 | PPD | Not Applicable – First Version |
| 2.0 | 21JUL2023 | PPD | Update the visit window for visit 5 following protocol amendment 3. SRT meetings to occur quarterly after all participants complete one-month post dose 2. SRC meetings on an ad-hoc basis. Changes following SRT and iSRC output review including percentages for solicited and unsolicited summaries to be out of the number of participants with a dose in each period update to the age categories and include summary for grade 2. Remove summaries for BMI, height and weight in the demography outputs. Updates to the estimands section. Include extra detail on the Deming's regression model. |
| 3.0 | 02FEB2024 | PPD | Include analysis of the duration of solicited events. Include the summary of the number of immunogenicity records to be imputed. Include immune concordance analysis. |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## **TABLE OF CONTENTS**

| 1. | LIST OF ABBREVIATIONS | 8 |
|---|---|---|
| 2. | INTRODUCTION | 11 |
| 3. | STUDY OBJECTIVES AND ESTIMANDS | 11 |
| 3.1. | Primary Objective | 11 |
| 3.2. | Secondary Objectives | 11 |
| 3.3. | Tertiary Objectives | 11 |
| 3.4. | Estimands | 11 |
| 4. | STUDY DESIGN | 19 |
| 4.1. | General Description | 19 |
| 4.2. | Schedule of Events | 22 |
| 4.3. | Changes to Analysis from Protocol | 22 |
| 5. | PLANNED ANALYSES | 22 |
| <b>5.1.</b> 5.1. | Data Monitoring Committee (DMC) | |
| 5.2. | Interim Analysis | 23 |
| 5.3. | Final Analysis | 24 |
| 6. | ANALYSIS SETS | 24 |
| 6.1. | Process for Analysis Set Assignment | 24 |
| 6.2. | Enrolled Set [ENR] | 25 |
| 6.3. | Exposed Set [ES] | 25 |
| 6.4. | Per Protocol Set [PPS] | 25 |
| Docur | hent: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\21374\(HPV9)\Biostatistics\Documentation\SAP\GSK_213749(HPV9-AS04-001)_WZA97329_SAP_Final_v3.0_02FEB2024.docx | 9 |
| Autho | or: PPD Version Number: | 3.0 |

Template No.: CS\_TP\_BS016 Revision 7

Reference: CS\_WI\_BS005

02FEB2024

Version Date:




#### Statistical Analysis Plan

| 7. | GENERAL CONSIDERATIONS | 26 |
|---|---|---|
| 7.1. | Reference Start Date and Study Day | 26 |
| 7.2. | Baseline | 26 |
| 7.3. | Retests, Unscheduled Visits and Early Termination Data | 27 |
| 7.4. | Windowing Conventions | 27 |
| 7.5. | Statistical Tests | 28 |
| 7.6. | Common Calculations | 28 |
| 7.7. | Software Version | 29 |
| 8. | STATISTICAL CONSIDERATIONS | 29 |
| 8.1. | Adjustments for Covariates and Factors to be Included in Analyses | 29 |
| 8.2. | Multicenter Studies | 30 |
| 8.3. | Missing Data | 30 |
| 8.4. | Examination of Subgroups | 30 |
| 9. | OUTPUT PRESENTATIONS | 30 |
| 10. | DISPOSITION AND WITHDRAWALS | 30 |
| 10.1. | Disposition | 31 |
| 10.2. | Protocol Deviations | 31 |
| | 2.1. Protocol Deviations Related to Study Conduct | |
| | 2.2. Protocol Deviations Related to Immunogenicity Analysis | |
| 11. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 32 |
| 12. | GENERAL MEDICAL HISTORY AND EXAMINATIONS | |
| 13. | PRIOR AND CONCOMITANT VACCINATIONS | |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

14.

15.



Effective Date: 01Nov2021


| <b>16.</b> IMMU | UNOGENICITY OUTCOMES | | . 34 |
|---|---|---|---|
| 16.1. Prima | ary Immunogenicity | | 3/ |
| | mary Immunogenicity Variables & Derivations | | |
| | ercurrent Event Handling and Data Imputation for Primary | | |
| 16.1.3. Pri | mary Analysis of Primary Immunogenicity Variables | minunogementy variable(s) | 34 |
| 10.1.5. 111 | mary marysis of filmary immunogementy variables | | 57 |
| 16.2. Secon | idary Immunogenicity | | 34 |
| | condary Immunogenicity Variables & Derivations | | |
| 16.2.1.1. | Anti-HPV IgG antibody concentration | | |
| 16.2.1.2. | Anti-HPV IgG antibody seroconversion and seropositivit | y rate | 35 |
| 16.2.1.3. | Anti-HPV neutralizing antibody titers | | 35 |
| 16.2.1.4. | Anti-HPV neutralizing antibody seroconversion and sero | positivity rate | 35 |
| 16.2.1.5. | Correlation between anti-HPV IgG antibody concentration | n and anti-HPV neutralizing antibody | , |
| titers | 35 | | |
| 16.2.2. Into | ercurrent Event Handling and Data Imputation for Seconda | ry Immunogenicity Variable(s) | 36 |
| 16.2.3. An | alysis of Secondary Immunogenicity Variables | | 36 |
| 16.2.3.1. | Anti-HPV IgG antibody concentration | | 36 |
| 16.2.3.2. | Anti-HPV IgG antibody seroconversion and seropositivit | y rate | 36 |
| 16.2.3.3. | Anti-HPV neutralizing antibody titers | ······ | 36 |
| 16.2.3.4. | Anti-HPV neutralizing antibody seroconversion and sero | positivity rate | 37 |
| 16.2.3.5. | Correlation between anti-HPV IgG antibody concentration | n and anti-HPV neutralizing antibody | , |
| titers | 37 | | |
| 16.2.4. Exp | ploratory Immunogenicity Variables | | 38 |
| 16.2.4.1. | Anti-HPV IgG antibody concentration between group ass | essment | 38 |
| 16.2.4.2. | Anti-HPV IgG antibody seroconversion rate | | |
| 16.2.4.3. | Anti-HPV neutralizing antibody titers between group asset | | |
| 16.2.4.4. | Anti-HPV neutralizing antibody seroconversion rate | | |
| 16.2.4.5. | Comparison of Anti-HPV IgG antibody concentration and | d Anti-HPV neutralizing antibody tite | rs 39 |
| CCI | | | |
| 16.4. Sensi | tivity Immunogenicity Variables & Derivations | | 40 |
| 17. <b>SAFE</b> | FY AND REACTOGENICITY OUTCOMES . | ••••• | . 41 |
| 17.1. Prima | ary Safety and Reactogenicity | | 41 |
| 17.1.1. Pri | mary Safety and Reactogenicity Variables & Derivations | | 41 |
| Document: \ | \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSm | ithKline\HP\/\213749 | |
| | HPV9)\Biostatistics\Documentation\SAP\GSK_213749(HP\ | | |
| | 001) WZA97329 SAP Final v3.0 02FEB2024.docx | | |
| | PD PD | Version Number: | 3.0 |
| Autilioi. | | V CI SIUIT INUITIDET. | ٠.٠ |
| | | Version Date: 02FEB20 | 24 |
| Template No.: | CS_TP_BS016 Revision 7 | Reference: CS_WI_BS005 | |
| - | | | |




| 17.1.2. Inter | current Event Handling and Data Imputation for Primary Efficacy Variable(s) | 42 |
|---|---|---|
| | ary Analysis of Primary Safety and Reactogenicity Variables | |
| | Solicited Events | |
| | Unsolicited Events | |
| | Serious Adverse Events | |
| 17.1.3.4. | Laboratory parameters outside Normal Range | 44 |
| 17.2. Second | ary Safety and Reactogenicity | 45 |
| 17.2.1. Seco | ndary Safety and Reactogenicity Variables & Derivations | 45 |
| | current Event Handling and Data Imputation for Secondary Safety and Reactogenicity | |
| 17.2.3. Anal | ysis of Secondary Safety and Reactogenicity Variables | 45 |
| | Solicited Events | 45 |
| | Unsolicited Events | 46 |
| 17.2.3.3. | Potential immune-mediated disease | 47 |
| 17.2.3.4. | Pregnancy | 47 |
| 17.3. Labora | tory Parameters | 47 |
| 18. DATA | NOT SUMMARIZED OR PRESENTED | 47 |
| 19. REFER | ENCES | 49 |
| | . PROGRAMMING CONVENTIONS FOR OUTPUTS | |
| IQVIA Output ( | Conventions | 50 |
| Dates & Times | | 50 |
| Spelling Format | | 50 |
| Presentation of ' | Treatment Groups | 50 |
| Presentation of \ | /isits | 51 |
| Listings | | 51 |
| APPENDIX 2 | . PARTIAL DATE CONVENTIONS | 53 |
| Almoniah C. B | in / Consortant Madientiess | 53 |
| Aigorium ior Pi | ior / Concomitant Medications: | 33 |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


#### 1. LIST OF ABBREVIATIONS

AE Adverse Event

AESI Adverse Event of Special Interest

ALT Alanine Aminotransferase

ANOVA Analysis of variance

AST Aspartate Aminotransferase

ATC Anatomical Therapeutic Chemical

BMI Body Mass Index

BUN Blood Urea Nitrogen

CD Cluster of Differentiation

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

CI

COVID-19 Coronavirus disease 2019

CSR Clinical Study Report

DMC Data Monitoring Committee

eCRF Electronic Case Report Form

ECL Electrochemiluminescence assay

ENR Enrolled Set

ES Exposed Set

GCP Good Clinical Practice

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




GMC Geometric Mean Concentration

GMT Geometric Mean Titer

HPV Human Papillomavirus

ICE Intercurrent Events

IgG Immunoglobulin G

IM Intramuscularly

iSRC internal Safety Review Committee

LLOQ Lower Limit Of Quantification

MedDRA Medical Dictionary for Regulatory Activities

PBNA pseudovirion-based neutralization assay

PD Protocol Deviation

PDMP Protocol Deviations Management Plan

pIMD Potential immune-mediated disease

PPS Per Protocol Set

PT Preferred Term

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SD Standard Deviation

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

TFL Table, Figures and Listing

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS TP BS016 Revision 7 Reference: CS WI BS005




ULOQ Upper Limit Of Quantification

WBC White Blood Cells

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## 2. Introduction

This Statistical Analysis Plan (SAP) describes the rules and conventions to be used in the presentation and analysis of immunogenicity and safety data for Protocol 213749 (HPV9-AS04-001). It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This SAP is based on protocol amendment 3, dated 8<sup>th</sup> June 2023.

### 3. STUDY OBJECTIVES AND ESTIMANDS

## 3.1. Primary Objective

The primary objectives are:

- to evaluate the safety and reactogenicity of GSK's investigational adjuvanted human papillomavirus (HPV) vaccine formulations
- to evaluate the immune response to GSK's investigational adjuvated HPV vaccine formulations.

## 3.2. Secondary Objectives

The secondary objectives are:

- To evaluate the safety and reactogenicity of GSK's investigational adjuvanted HPV vaccine formulations
- To evaluate the immune response for all HPV vaccine types for all vaccines

# 3.3. Tertiary Objectives



#### 3.4. Estimands

The primary and secondary estimands to support regulatory decisions are described in the following table:

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021




### **Table A:** Objectives and Estimands

| Estimand | d Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment | Population | Variable (or | Intercurr | ent events (ICEs) | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| Primary | Randomized HPV dose (High, Medium or Low) or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Each grade 3 solicited<br>administration site<br>event within 7 days<br>after each vaccine<br>dose | 1. eDiary not<br>completed on each<br>day | 1. Missing data won't be imputed. All data collected will be included in the summaries (treatment policy). | Percentage of participants with event with exact 95% Confidence Interval (CI) |
| Primary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Each grade 3 solicited systemic event within 7 days after each vaccine dose | 1. eDiary not<br>completed on each<br>day | 1. Missing data won't be imputed. All data collected will be included in the summaries (treatment policy). | Percentage of participants with event with exact 95% CI |
| Primary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or Gardasil 9 | Female participants<br>between 16 and 26<br>years old | Each grade 3<br>unsolicited adverse<br>event within 28 days<br>after each vaccine<br>dose | 1. Permanently discontinuation from study treatment due to any reasons | 1. Missing data won't be imputed. All data collected will be included in the summaries (treatment policy). | Percentage of participants with event with exact 95% CI |
| Primary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Serious Adverse<br>Events from first<br>vaccination up to<br>study end | 1. Permanently discontinuation from study treatment due to any reasons | 1. Missing data won't be imputed. All data collected will be included in the summaries (treatment policy). | Percentage of participants with event with exact 95% CI |

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment | Population | Variable (or | Intercurre | ent events (ICEs) | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| Primary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or Gardasil 9 | Female participants<br>between 18 and 26<br>years old | Clinically relevant<br>abnormalities in each<br>biochemical and<br>hematological<br>parameter at Day 7<br>post-dose 1 | 1. Permanently discontinuation from study treatment due to any reasons | 1. Missing data won't be imputed. All data collected will be included in the summaries (treatment policy). | Percentage of participants in<br>Step 1 with event with exact<br>95% CI |
| Primary | Randomized HPV dose (High, Medium or Low) or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Anti-HPV immunoglobulin G (IgG) antibody 1 month after third dose (Month 7) | 1. Permanently discontinuation from study treatment due to any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood sample taken out of window 5. No post-vaccine immunogenicity result available | 1. Missing data won't be imputed. 2. Participant excluded from the immunogenicity analysis. 3. Participant excluded from the immunogenicity analysis. 4. Participant excluded from the immunogenicity analysis. 5. Participant excluded from the immunogenicity analysis. | Antibody GMC with exact 95% CI. |
| Secondary | Randomized HPV dose (High, | Female participants between 16 and 26 | Each solicited administration site | 1. eDiary not completed on each | 1. Missing data won't be imputed. All data | Percentage of participants with event with exact 95% CI |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | | | | Attributes | | |
|---|---|---|---|---|---|---|
| | Treatment | Population | Variable (or | Intercurr | ent events (ICEs) | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| | Medium or Low) or Gardasil 9 | years old | event within 7 days | day | collected will be included in the summaries | |
| | of Garaasti 9 | | dose | | (treatment policy). | |
| Secondary | Randomized HPV | Female participants | Each solicited | 1. eDiary not | 1. Missing data won't be | Percentage of participants with |
| | dose (High, | between 16 and 26 | systemic event within | completed on each | imputed. All data | event with exact 95% CI |
| | Medium or Low) | years old | 7 days after each | day | collected will be included | |
| | or Gardasil 9 | | vaccine dose | | in the summaries (treatment policy). | |
| Secondary | Randomized HPV | Female participants | Unsolicited adverse | 1. Permanently | 1. Missing data won't be | Percentage of participants with |
| , | dose (High, | between 16 and 26 | event within 28 days | discontinuation | imputed. All data | event with exact 95% CI |
| | Medium or Low) | years old | after each vaccine | from study | collected will be included | |
| | or Gardasil 9 | | dose | treatment due to | in the summaries | |
| | | | | any reasons | (treatment policy). | |
| Secondary | Randomized HPV | Female participants | Potential immune- | 1. Permanently | 1. Missing data won't be | Percentage of participants with |
| | dose (High, | between 16 and 26 | mediated disease | discontinuation | imputed. All data | event with exact 95% CI |
| | Medium or Low) | years old | (pIMDs) from first | from study | collected will be included | |
| | or Gardasil 9 | | vaccination up to | treatment due to | in the summaries | |
| | | | study end | any reasons | (treatment policy). | |
| Secondary | Randomized HPV | Female participants | Experienced | 1. Permanently | 1. Missing data won't be | Percentage of participants who |
| | dose (High, | between 16 and 26 | pregnancy and their | discontinuation | imputed. All data | experienced pregnancy and their |
| | Medium or Low) | years old | outcomes from Day 1 | from study | collected will be included | outcomes |
| | or Gardasil 9 | | of pregnancy up to | treatment due to | in the summaries | |
| | | | study end | any reasons | (treatment policy). | |
| Secondary | Randomized HPV | Female participants | Anti-HPV IgG | 1. Permanently | 1. Missing data won't be | Antibody GMC and 2-sided 95% |
| | dose (High, | between 16 and 26 | antibody | discontinuation | imputed. | CI at each timepoint. GMC ratio |
| | Medium or Low) | years old | concentration at Day | from study | 2. Participant excluded | at Month 3 and Month 7 |
| | or Gardasil 9 | | 1, Month 2, Month 3, | treatment due to | from the immunogenicity | |

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | d Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment Population Variable (or Intercurrent events (ICEs) | | | | | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| | | | Month 6, Month 7<br>and Month 12 | any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood sample taken out of window 5. No post-vaccine immunogenicity result available | analysis. 3. Participant excluded from the immunogenicity analysis. 4. Participant excluded from the immunogenicity analysis. 5. Participant excluded from the immunogenicity analysis. | |
| Secondary | Randomized HPV dose (High, Medium or Low) or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Anti-HPV IgG<br>antibody<br>seroconversion at<br>Month 2, Month 3,<br>Month 6, Month 7<br>and Month 12 | 1. Permanently discontinuation from study treatment due to any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood | Missing data won't be imputed. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity | Seroconversion and seropositivity rates for each antigen with exact 95% CI. Difference in seroconversion rate at Month 3 and Month 7 with exact 95% CI. |

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment | | | Intercurre | ent events (ICEs) | Population level summary |
| | | | endpoint) | Description | Handling strategy | 7 |
| | | | | sample taken out of window 5. No post-vaccine immunogenicity result available | analysis. | |
| Secondary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or Gardasil 9 | Female participants<br>between 16 and 26<br>years old | Anti-HPV neutralizing antibody titers at Day 1, Month 3 and Month 7 (at least 150 participants in each group) and Month 2 in a subset of participants | 1. Permanently discontinuation from study treatment due to any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood sample taken out of window 5. No post-vaccine immunogenicity result available | 1. Missing data won't be imputed. 2. Participant excluded from the immunogenicity analysis. 3. Participant excluded from the immunogenicity analysis. 4. Participant excluded from the immunogenicity analysis. 5. Participant excluded from the immunogenicity analysis. | Antibody Geometric Mean Titer (GMT) with exact 95% CI at each timepoint and GMT ratio at Month 3 and Month 7. |
| Secondary | Randomized HPV dose (High, Medium or Low) or <i>Gardasil 9</i> | Female participants<br>between 16 and 26<br>years old | Anti-HPV<br>neutralizing antibody<br>seroconversion at<br>Month 3 and Month 7 | 1. Permanently discontinuation from study treatment due to | Missing data won't be imputed. Participant excluded from the immunogenicity | Seroconversion and seropositivity rates for each antigen with exact 95% CI. Difference in seroconversion |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | Attributes Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment | Population | Variable (or | Intercurrent events (ICEs) | | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| | | | | any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood sample taken out of window 5. No post-vaccine immunogenicity result available | analysis. 3. Participant excluded from the immunogenicity analysis. 4. Participant excluded from the immunogenicity analysis. 5. Participant excluded from the immunogenicity analysis. | rate at Month 3 and Month 7 with exact 95% CI. |
| Secondary | Randomized HPV<br>dose (High,<br>Medium or Low)<br>or Gardasil 9 | Female participants<br>between 16 and 26<br>years old | anti-HPV IgG<br>antibody<br>concentration and<br>anti-HPV neutralizing<br>antibody titers at Day<br>1, Month 2, Month 3<br>and Month 7 | 1. Permanently discontinuation from study treatment due to any reasons 2. Study vaccine not administered per protocol 3. Prohibited medication or intercurrent medical condition 4. Vaccine or blood | Missing data won't be imputed. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity analysis. Participant excluded from the immunogenicity | Correlation between anti-HPV IgG antibody concentration and anti-HPV neutralizing antibody titers for each timepoint. Functional relationship between each pair of assay methods. A qualitative summary between ECL and PBNA for each timepoint. |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021



Statistical Analysis Plan


| Estimand | Attributes | | | | | |
|---|---|---|---|---|---|---|
| | Treatment | Population | Variable (or | Intercurrent events (ICEs) | | Population level summary |
| | | | endpoint) | Description | Handling strategy | |
| | | | | sample taken out of | analysis. | |
| | | | | window | | |
| | | | | 5. No post-vaccine | | |
| | | | | immunogenicity | | |
| | | | | result available | | |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021


#### 4. STUDY DESIGN

## 4.1. General Description

This is a phase 1/2 randomized, observer-blind, multi-country study with 4 groups of females 16-26 years of age at the time of vaccine administration. Participants will be randomized in a 1:1:1:1 ratio to receive a series of 3 investigational adjuvanted intervention doses (3 different potencies [a high, medium, low potency]) or a series of the *Gardasil 9* vaccine.

The investigational adjuvanted intervention or *Gardasil 9* vaccine will be administered intramuscularly (IM) at Day 1 (Month 0), Month 2, and Month 6. Blood sampling will be performed on Day 1, Month 2, Month 3, Month 6, Month 7, and Month 12 to assess for immunological response.

This study is organized into 2 steps. Forty-eight participants (12 per group) of the study Step 1 (sentinel participants) will receive the initial assigned dose prior to participants in Step 2 of the study, and sentinel participants will have an additional blood sampling visit at Day 7 to assess for biochemical and hematological parameters. The internal Safety Review Committee (iSRC) will review the accumulated safety data up to 7 days post-dose 1 for the sentinel participants to determine whether any of the pre-defined holding rules have been met. If no safety concerns were observed and no holding rules were met, the sentinel participants will continue with study visits and dosing as scheduled, and the Step 2 participants will be initiated.



Approximately 1080 participants will be randomly assigned to the 4 study groups to provide approximately 270 participants per study group.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




### **Table B:** Study intervention Groups

| Study Group | Study Interventions | Number of Participants |
|-------------|---------------------|------------------------|
| HPV9High | HPV9-High | 270 |
| HPV9Med | HPV9-Medium | 270 |
| HPV9Low | HPV9-Low | 270 |
| Gar9 | Gardasil 9 | 270 |

The duration of the intervention will be approximately 6 months. Participants will be monitored until Month 12. Monitoring of pregnancies (if any) can be beyond 12 months.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


3.0

02FEB2024

Version Number: Version Date:

#### Figure 1 Study Design Overview



Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Author:

PPD




&iSRC reviews Sentinel participants post-dose 1 safety data, then iSRC reviews the data on monthly basis until one month post-dose 2 for all participants and one-month post dose 3 for Step 1 participants are reviewed Safety data review will occur then on a quarterly basis till the end of the study.

%Blood sampling for biochemistry and hematology is only for Step 1 participants.

#### 4.2. Schedule of Events

Schedule of events can be found in Table 1 of the protocol.

## 4.3. Changes to Analysis from Protocol

- Differences in the seroconversion rates between study groups are to be summarized for the anti-HPV IgG
   Antibody and the anti-HPV Neutralizing Antibody
- Sensitivity analysis of the anti-HPV IgG Antibody and the anti-HPV Neutralizing Antibody included where the values above the Upper Limit of Quantification (ULOQ) are not imputed.

## 5. PLANNED ANALYSES

The following analyses will be performed for this study:

- Analyses for iSRC review
- Two Interim Analyses
- Final Analysis

# 5.1. Data Monitoring Committee (DMC)

Safety monitoring review will be performed by the iSRC.

#### 5.1.1. iSRC review

An iSRC will be reviewing the unblinded accumulated safety data up to 7 days post-dose 1 for the sentinel participants to determine whether any of the pre-defined holding rules have been met in order to proceed with study schedule of activities. Then iSRC will review the safety data on a monthly basis until safety data from one-month

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




post-dose 2 for all participants and data from one-month post dose 3 for Step 1 participants are reviewed. The iSRT will then review the safety data on a quarterly basis until the end of the study. Further details on this analysis will be provided in a separate analysis plan.

## 5.2. Interim Analysis

Two interim analyses will take place for this study.

The first will be performed on all data available for the primary and secondary endpoints up to Month 3 (1 month post-dose 2). This includes all safety data up to 1-month post-dose 2 for all participants, anti-HPV IgG data up to 1-month post-dose 2 for all participants\* and anti-HPV neutralizing titers data up to 1-month post-dose 2 with at least 150\* participants/group for 1-month post-dose 2 timepoint. Unblinded analysis will also be provided with the study groups unblinded, no individual unblinding information will be shared. Listings will be provided in a blinded manner. Summary analysis might lead to accidental unblinding.

The second will be performed on all available data for primary and secondary endpoints up to Month 7 (1 month post-dose 3). This includes all safety data up to 1-month post-dose 3 for all participants, anti-HPV IgG data up to 1-month post-dose 3 for all participants and anti-HPV neutralizing titers data up to 1-month post-dose 3 with at least 150\* participants/group for 1-month post-dose 3 timepoint. Unblinded analysis will also be provided with the study groups unblinded, no individual unblinding information will be shared. Listings will be provided in a blinded manner. Summary analysis might lead to accidental unblinding.

\*In case of visit delay, analysis may be performed for as many participants as possible with data available at the time of the analysis. Analysis for remaining participants will be performed at the time of the next analysis.

The results of these will be based on the unblinded treatment groups. See section 9.5 of the protocol for more details.

Derivations and definitions for the interim analysis will be based on those required for the final analysis contained in this analysis plan unless deviations are stated within the text. The list of outputs provided with the full set of output templates (planned for the final analysis) will highlight which of these outputs will also be provided for the interim analysis.

The IQVIA study team, including those responsible for creating the programs to produce the outputs for the Interim

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




Analysis, will remain blinded. Once the programs have been produced by the IQVIA study team, these programs will be sent to an independent statistician who will apply the randomization schedule and provide a set of unblinded outputs.

## 5.3. Final Analysis

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics following Sponsor Authorization of this Statistical Analysis Plan, Database Lock, Sponsor Authorization of Analysis Sets and Unblinding of intervention group.

This SAP is focused/limited to planned interim and final analyses. Outputs required for the interim analyses will be flagged in the Table, Figures and Listings (TFL) mock shells document.

### 6. ANALYSIS SETS

Agreement and authorization of subjects included/excluded from each analysis set will be conducted prior to the unblinding of the study.

## 6.1. Process for Analysis Set Assignment

- Definitions for analysis sets are provided below.
- Prior to database lock, a transfer of raw data from the electronic Case Report Form (eCRF) will occur, and
  participants will be assigned to analysis sets in accordance with the definitions in this SAP and the available
  data at that time. However, the protocol deviations will be monitored continuously throughout the study.
- Listings presenting participants excluded from each preliminary analysis set and reasons for exclusion will be
  prepared for sponsor review ahead of database lock in order to allow appropriate related data queries to be
  issued.
- Listings presenting participants excluded from each final analysis set and reasons for exclusion will be prepared
  for sponsor review ahead of unblinding for a final review and approval. However, for deviations that can only
  be assessed after unblinding such as vaccination errors these will be reviewed after unblinding.
- A Data Review meeting will be held to confirm analysis set assignment for each participant and any changes
  will be recorded. Changes will be implemented, and an updated analysis set assignment will be approved by the
  sponsor.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




- Sponsor authorization of the analysis sets will be necessary to unblind the data after the final database lock.
   Once approved, the study will be unblinded, analysis sets will be finalized including additional eliminations requiring unblinding, and the database will be locked.
- After database lock, the final analysis sets will be derived using the final study data, i.e., clinical database (eCRF), external vendor data (immunogenicity results), protocol deviations log and blinded data report.

## 6.2. Enrolled Set [ENR]

All eligible participants who received a study vaccine or had a blood draw before study vaccine administration or were randomized. Note that as per Good Clinical Practice (GCP) enrolled participants should have completed the informed consent process and participants should be eligible before initiating any study procedure.

## 6.3. Exposed Set [ES]

All participants who received a study intervention. Analysis per group is based on the study vaccine administered

## 6.4. Per Protocol Set [PPS]

A per-protocol set (PPS) will be defined for all participants in the ES at each visit that meet the following criteria:

- Meeting all eligibility criteria
- For whom the administration route of the vaccine was as according to protocol
- For whom the study vaccine was administered per protocol
- Who did not receive a concomitant medication/product/vaccine leading to exclusion from a PP analysis, as
  described in the protocol
- Who did not present with an intercurrent medical condition leading to exclusion from a PP analysis, as described in the protocol
- Who complied with the vaccination schedule
- Who complied with the timings of the post-vaccination blood sampling for immune response evaluation
- For whom post-vaccination immunogenicity results are available for at least one antigen at the corresponding time points

The eliminations for the PPS will be adapted as per the timepoint analysis, e.g., for month 3 analysis only violations up to month 3 will be excluded.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


#### 7. GENERAL CONSIDERATIONS

Data will be summarized descriptively (frequency and percentage for categorical data and mean, standard deviation [SD] and range for continuous data, unless specified otherwise). In summary tables for categorical data for which categories are defined on the eCRF, all categories will be presented as specified, even if the participant count within that category is zero.

Unless otherwise specified, all data collected during the trial will be presented in listings for the ENR.

## 7.1. Reference Start Date and Study Day

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of the most recent dose of study vaccination and will appear in every listing where an assessment date or event date appears.

If the date of the event is on or after the date of vaccination then:

Study Day = (date of event – date of vaccination) + 1.

If the date of the event is prior to the date of vaccination then:

Study Day = (date of event – date of vaccination).

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

#### 7.2. Baseline

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered baseline if the assessment is planned per protocol to take place prior to first study vaccination administration. Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline unless otherwise indicated based on available start date/time

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


combination or collected eCRF information that identifies the individual event/medication as starting prior to first study vaccination administration.

## 7.3. Retests, Unscheduled Visits and Early Termination Data

In general, for by-visit summaries, data recorded at the nominal visit will be presented. Unscheduled measurements will not occur for this study.

Listings will include all scheduled, and early termination discontinuation data.

# 7.4. Windowing Conventions

Allowed time window for each visit will be performed as mentioned in "Schedule of Activities", section 1.3 of protocol.

**Table C:** Intervals Between Study Visits

| Interval | Planned Visit Interval* | Allowed Interval Range |
|---|---|---|
| Visit 1 → Visit 2 | 7 days | 7 – 12 days |
| Visit 1 → Visit 3 | 60 days | 56 – 74 days |
| Visit 3 → Visit 4 | 28 days | 28 – 44 days |
| Visit 1 → Visit 5 (visit 5 occurring before protocol amendment 2 [08JUN2023]) | 180 days | 180 – 194 days |
| Visit 1 → Visit 5 (visit 5 occurring on or after protocol amendment 2 [08JUN2023]) | 180 days | 166 – 194 days |
| Visit 5 → Visit 6 | 28 days | 28 – 44 days |
| Visit 1 → Visit 7 | 360 days | 346 – 374 days |

<sup>• \* =</sup> Number of days between the visits

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


**Table D:** Window Convention

| Assigned Study Day | Visit Label as per Protocol | Visit Assigned |
|---|---|---|
| Day 1 | Visit 1 | Visit 1 |
| Day 7 (Day 1 + 7 to 12 days) | Visit 2 | Visit 2 |
| Day 60 (Day 1 + 56 to 74 days) | Visit 3 | Visit 3 |
| Day 88 (Day 1 + 84 to 118 days) | Visit 4 | Visit 4 |
| Day 180 (Day 1 + 180 to 194 days) (visit 5 occurring before protocol amendment 2 [08JUN2023]) | Visit 5 | Visit 5 |
| Day 180 (Day 1 + 166 to 194 days) (visit 5 occurring on or after protocol amendment 2 [08JUN2023]) | Visit 5 | Visit 5 |
| Day 208 (Day 1 + 208 to 238 days) | Visit 6 | Visit 6 |
| Day 360 (Day 1 + 346 to 374 days) | Visit 7 | Visit 7 |

#### 7.5. Statistical Tests

The default significant level will be 5%; CIs will be 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

#### 7.6. Common Calculations

Geometric Mean Concentration/Titer (GMC/GMT):

Distributions of antibodies are generally skewed to the right (Nauta, 2010). Therefore, prior to any statistical analysis that assumes normally distributed observations, antibody concentrations or titers will be log10-transformed. GMC/GMTs and their 95% CI are computed by exponentiating (base 10) the least squares mean and 95% CI of the log10 titers.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




The GMC/GMT will be calculated using the following formula:

$$10^{\left(\frac{\sum_{i=1}^{n}\log 10(t_i)}{n}\right)}$$

Where  $t_1, t_2, ..., t_n$  are n observed immunogenicity concentrations/titer.

Concentration below assay cut-off (i.e., <lower limit of quantification or < LLOQ) will be replaced by half the assay cut-off (LLOQ/2) for the purpose of GMC computation. Any concentrations above the upper limit of quantification (or ULOQ) will be set to the ULOQ value. No imputation for ULOQ will be performed for the sensitivity analysis of GMC/GMT and for the correlations and Deming's regression.

#### Seroconversion:

Defined as the appearance of antibodies (i.e., concentrations/titers greater than or equal to the cut-off value) in the serum of participants seronegative before vaccination.

For quantitative measurements, change from baseline will be calculated as:

• Test Value at Visit X – Baseline Value

#### 7.7. Software Version

All analyses will be conducted using SAS version 9.4 or higher.

#### 8. STATISTICAL CONSIDERATIONS

# 8.1. Adjustments for Covariates and Factors to be Included in Analyses

For details on the factors to be used in the analysis refer to section 17.1 and 17.2. The model will include all groups and country as fixed categorical effects in the ANOVA model.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


### 8.2. Multicenter Studies

This study will be conducted by multiple investigators at multiple centers. The participants will be randomized to one of the 4 groups (refer to Table B in section 4.1) which will be performed in a 1:1:1:1 ratio prior to intervention to provide approximately 270 enrolled participants per group.

## 8.3. Missing Data

Missing data (missing, incomplete, or partial dates, AE measurement (including missing AE severity and relationship), prior and concomitant medications and death date) will be handled as per APPENDIX 2 of this analysis plan.

Missing immunogenicity data will not be imputed.

## **8.4.** Examination of Subgroups

No subgroup analyses will be performed for this study.

## 9. OUTPUT PRESENTATIONS

APPENDIX 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics. Statistical output numbering will follow 'ICH E3 Structure and Content of Clinical Study Reports'.

#### 10. DISPOSITION AND WITHDRAWALS

All participants who are enrolled in the study (those who received a study intervention or were randomized) will be accounted for in this study.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




## 10.1. Disposition

Participant disposition, withdrawals, and reasons for exclusion from each analysis set, including inclusion as well as exclusion criteria will be presented for the ENR. Specifically, the number of participants, vaccinated, completed the study, discontinuing the study and the reason for discontinuation will be summarized by study group for the ENR. Additionally, the number of participants returning for each visit for the ES will be presented. The number of participants enrolled by age category (preterm newborn – gestational age < 37 weeks, newborn (0-27 days), infant and toddler (28 days to 23 months), children (2-11 years), adolescents (12-17 years), 18-64 years, 65-84 years and >=85 years) will be summarized by study group.

A listing of the disposition for all participants with early withdrawal or discontinuation due to having Coronavirus Disease 2019 (COVID-19) or COVID-19 related issues information will be provided. The number of participants who discontinue the study due to COVID-19 will also be summarized by study group.

#### **10.2.** Protocol Deviations

During the study, Protocol Deviations (PDs) will be collected in a PD log, as detailed in the Protocol Deviations Management Plan (PDMP). All PDs will be assessed as either important or non-important. PDs will be reviewed by the sponsor, and their status confirmed by the time that all data are cleaned for the Final Analysis. A summary table presenting the number and percentage of participants with important PDs (i.e, those PDs associated to elimination from PPS) will be presented for participants in the ES. A listing of all PDs including an indicator of those excluded from the PPS and an indicator of COVID-19 causality will be provided.

#### 10.2.1. Protocol Deviations Related to Study Conduct

A PD is any non-compliance with the clinical trial protocol, GCP, or protocol deviation guidelines requirements. The non-compliance may be either on the part of the participant, the site investigator, the study site staff or the sponsor.

### 10.2.2. Protocol Deviations Related to Immunogenicity Analysis

Changes to the procedures or events, which may impact the quality of the immunogenicity data, will be considered important PDs and will be described within the Clinical Study Report (CSR). This includes any circumstances that

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

\_\_\_\_\_


could alter the evaluation of the immunogenicity results such as sample processing errors that lead to inaccurate immunogenicity results, and/or inaccurate dosing which could exclude them from the PPS. In addition, participants may also be eliminated from the PPS based on usage of certain concomitant therapies or vaccines as described in Section 5.2.2 of the Protocol.

### 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the ES and each of the PPS. No statistical testing will be carried out for demographic or other baseline characteristics. The following demographic and other baseline characteristics will be reported for this study:

- Age (years) calculated relative to date of first vaccination
- Age category -<18 and >=18
- Race (as per Clinical Data Interchange Standards Consortium [CDISC] categories)
- Ethnicity

## 12. GENERAL MEDICAL HISTORY AND EXAMINATIONS

Medical/Vaccination History information will be presented for the ENR.

- Medical History will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, Version 26.0 or higher.
- Data captured on the "Medical History" page of the eCRF will be presented by System Organ Class (SOC) and Preferred Term (PT). Medical occurrences that begin before the start of study intervention but after obtaining informed consent will be recorded on the Medical History section of the eCRF, not the AE section.

Data will be presented in table summaries for general medical/vaccination history for the ENR and in listings.

### 13. PRIOR AND CONCOMITANT VACCINATIONS

Prior and concomitant and co-administered vaccination will be coded with the current version of the WHO drug dictionary.

• Prior vaccinations are vaccinations per protocol given to participants prior to the dosing of study intervention and are recorded on the eCRF.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




• Concomitant vaccinations are defined as any vaccine that the participant is receiving as of the time of enrolment or receives during the study (other than study interventions) as recorded on the "Concomitant Medications/Vaccination" page of the eCRF, under the "Concomitant Vaccination" category.

Data will be presented in table summaries for concomitant vaccinations for the ES and in listings.

### 14. MEDICATIONS

The percentage of participants who started medications after study vaccination will be presented by intervention group for the ES.

See APPENDIX 2 for handling of partial dates for medications, in the case where it is not possible to define a medication as prior or concomitant, the medication will be classified by the worst case; i.e., concomitant.

- 'Prior' medications are medications which started prior to the dose of study vaccination.
- 'Concomitant' medications are medications which started on or after the day of the administration of study vaccination

Further details are in Section 6.8 of the Protocol. Concomitant medications during the study will be presented in table summaries (Any, any antipyretic, any prophylactic antipyretic, any antibiotic) and in listings for all medications.

## 15. STUDY VACCINATION EXPOSURE

Exposure to study vaccine will be presented for the ES. Summaries will include the number of participants with exactly 1 dose, exactly 2 doses, exactly 3 doses, at least 1 dose and at least 2 doses. The date and time of study vaccine administration will be taken from the eCRF "Exposure" form. For dosing instructions and route, refer to Table 6 of the Protocol.

Data will also be presented in listings.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## 16. IMMUNOGENICITY OUTCOMES

## 16.1. Primary Immunogenicity

#### 16.1.1. Primary Immunogenicity Variables & Derivations

The primary immunogenicity endpoint is:

• Anti-HPV immunoglobulin G (IgG) antibody geometric mean concentrations (GMCs), 1 month after the third dose (Month 7) for each antigen. For the derivation of GMC refer to section 7.6.

# 16.1.2. Intercurrent Event Handling and Data Imputation for Primary Immunogenicity Variable(s)

See Table A: and section 8.3.

#### 16.1.3. Primary Analysis of Primary Immunogenicity Variables

The primary immunogenicity analysis will be performed for the PPS. If the number of participants excluded from the PPS is >5% when compared with the ES, then the analysis will also be performed for the ES.

The primary immunogenicity endpoint GMCs of anti-HPV IgG antibody concentration at Month 7 will be summarized by study group for each antigen with their 95% CI summarised for the pre-vaccination status of seronegative, seropositive and total. Anti-HPV IgG antibody concentration will be graphically presented by reverse cumulative curves per study group.

# 16.2. Secondary Immunogenicity

The secondary immunogenicity analyses will be performed for the PPS.

#### 16.2.1. Secondary Immunogenicity Variables & Derivations

#### 16.2.1.1. ANTI-HPV IGG ANTIBODY CONCENTRATION

Anti-HPV IgG antibody concentration at Day 1, Month 2, Month 3, Month 6, and Month 12 for each antigen.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




#### 16.2.1.2. ANTI-HPV IGG ANTIBODY SEROCONVERSION AND SEROPOSITIVITY RATE

Anti-HPV IgG antibody seroconversion and seropositivity rates at Day 1 (for seropositivity only), Month 2, Month 3, Month 6, Month 7 and Month 12 for each antigen.

Seroconversion is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the cut-off value) in the serum of participants seronegative before vaccination.

Seropositivity is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the cut-off value) in the serum of participants.

#### 16.2.1.3. ANTI-HPV NEUTRALIZING ANTIBODY TITERS

Anti-HPV neutralizing antibody titers at Day 1, Month 3 and Month 7 (at least 150 participants in each group) and Month 2 in a subset of 384 participants (at least 96 in each group) for each antigen.

16.2.1.4. ANTI-HPV NEUTRALIZING ANTIBODY SEROCONVERSION AND SEROPOSITIVITY RATE Anti-HPV neutralizing antibody seroconversion and seropositivity rates at Day 1 (seropositivity only), Month 3 and Month 7 (at least 150 participants in each group) and Month 2 in a subset of 384 participants (at least 96 in each

group) for each antigen.

Seroconversion is defined as the appearance of antibodies (i.e, titer greater than or equal to the cut-off value) in the serum of participants seronegative before vaccination.

Seropositivity is defined as the appearance of antibodies (i.e, titer greater than or equal to the cut-off value) in the serum of participants.

16.2.1.5. CORRELATION BETWEEN ANTI-HPV IGG ANTIBODY CONCENTRATION AND ANTI-HPV NEUTRALIZING ANTIBODY TITERS

Correlation between anti-HPV IgG antibody concentrations and anti-HPV neutralizing antibody titers at Day 1, Month 2, Month 3, Month 7 and overall for each antigen.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



## 16.2.2. Intercurrent Event Handling and Data Imputation for Secondary Immunogenicity Variable(s)

See Table A: and section 8.3.

## 16.2.3. Analysis of Secondary Immunogenicity Variables

#### 16.2.3.1. ANTI-HPV IGG ANTIBODY CONCENTRATION

The immunogenicity endpoint GMCs of anti-HPV IgG antibody concentration will be summarized for each antigen at Day 1, Month 2, Month 3, Month 6, and Month 12 by study group with their 95% CI derived considering log10-transformed antibody concentrations are normally distributed with unknown variance, summarised for the prevaccination status of seronegative, seropositive and total. The concentration below the assay cut-off will be assigned to half the cut-off for the purpose of GMC computation. The number of records above the ULOQ will be summarised at each visit for the pre-vaccination status of seronegative (except Day 1), seropositive and total.

Anti-HPV IgG antibody concentration will be graphically presented by reverse cumulative curves per antigen, timepoint and study group.

#### 16.2.3.2. ANTI-HPV IGG ANTIBODY SEROCONVERSION AND SEROPOSITIVITY RATE

The percentage of participants with a seroconversion and seropositivity for each antigen will be summarized for each antigen at Day 1 (for seropositivity only), Month 2, Month 3, Month 6, Month 7 and Month 12 by study group and corresponding 2-sided 95% CI will be reported based on Clopper and Pearson method.

## 16.2.3.3. ANTI-HPV NEUTRALIZING ANTIBODY TITERS

The anti-HPV neutralizing antibody titers will be summarized for each antigen at Day 1, Month 3 and Month 7 (at least 150 participants in each group) and Month 2 in a subset of participants by study group with their 95% CI derived considering log10-transformed antibody titers are normally distributed with unknown variance, summarised for the pre-vaccination status of seronegative, seropositive and total. Anti-HPV neutralizing antibody titers will be graphically presented by reverse cumulative curves per antigen, timepoint and study group. The concentration below the assay cut-off will be assigned to half the cut-off for the purpose of GMT computation. The number of records above the ULOQ will be summarised at each visit for the pre-vaccination status of seronegative (except day 1), seropositive and total.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Telephone Telephone English Telephone English




## 16.2.3.4. ANTI-HPV NEUTRALIZING ANTIBODY SEROCONVERSION AND SEROPOSITIVITY RATE

The percentage of participants with a seroconversion and seropositivity for each antigen will be summarized at Day 1 (seropositivity only), Month 3 and Month 7 and Month 2 in a subset of 384 participants (at least 96 in each group) by study group and corresponding 2-sided 95% CI will be reported based on Clopper and Pearson method.

## 16.2.3.5. CORRELATION BETWEEN ANTI-HPV IGG ANTIBODY CONCENTRATION AND ANTI-HPV NEUTRALIZING ANTIBODY TITERS

The Pearson coefficient of correlation between anti-HPV IgG antibody concentration and anti-HPV neutralizing antibody titers with associated p-value will be calculated for each investigational adjuvanted vaccine groups and *Gardasil 9* group for each antigen at Day 1, Month 2, Month 3, Month 7 and overall. The Pearson correlation will be computed by the log10-transformation of specific antibody concentrations.

For each HPV type, the functional relationship between the pair of assay methods (pseudovirion-based neutralization assay [PBNA] verses electrochemiluminescence assay [ECL]) will be estimated by timepoint at Day 1, Month 2, Month 3 and Month 7 and overall using the Deming's regression model.

The Deming's regression will consider the following:

- Anti-HPV Neutralizing titers (from PBNA) with errors  $\epsilon_i$
- 1.1  $x_i = X_i + \epsilon_i$ 
  - Anti-HPV IgG antibody concentrations (from ECL) with errors  $\delta_{ij}$
- 1.2  $y_i = Y_i + \delta_i$

where X<sub>i</sub> and Y<sub>i</sub> are the measurements of Anti-HPV Neutralizing titers and Anti-HPV IgG antibody concentrations.

The Deming's regression model to be fitted is

$$Y = \beta_0 + \beta_1 X$$

The following terms will be fitted in the model:

Response (Y): log transformed anti-HPV IgG antibody concentration (from ECL)

Covariate (X): log transformed anti-HPV Neutralizing titers (from PBNA)

 $\beta_0$  is the Y-intercept and  $\beta_1$  is the coefficient (slope) associated with the Anti-HPV Neutralizing titers from PBNA.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




Assumption: Error ratio:  $V(\epsilon_i) / V(\delta_i) = 1$ 

The model will be fitted for each antigen and study group separately.

The intercept and the slope estimates and corresponding 95% CI (only for slope) will be presented. Note that a slope  $\approx$  1 implies a favorable outcome, i.e. both the assays (ECL and PBNA) are in strong agreement and have a similar performance.

Graphs representing the scatterplot of the Anti-HPV Neutralizing titers and Anti-HPV IgG antibody concentration will be presented for all timepoints with the Deming's regression line for each antigen and each study group. LLOQ and ULOQ values of the ECL and PBNA will also be presented in the same graph.

#### 16.2.4. **Exploratory Immunogenicity Variables**

The exploratory immunogenicity analyses will be performed for the Month 3 and Month 7 PPS.

16.2.4.1. ANTI-HPV IGG ANTIBODY CONCENTRATION BETWEEN GROUP ASSESSMENT Anti-HPV IgG antibody concentration at Month 3 and Month 7 for each antigen.

For each antigen an adjusted GMC and GMC ratio with 2-sided 95% CI for intervention group which is derived from an ANOVA model on log10 transformed concentration will be tabulated for anti-HPV IgG antibody concentration adjusted for country effect. The analysis will be performed at Month 3 and at Month 7, summarised for the pre-vaccination status of seronegative, seropositive and total. The model will be based on the data from all groups, will include study group and country as a fixed effect and will be based on the PPS. The non-inferiority of different vaccine formulations to the control group will be assessed if the lower limit of the 2-sided 95% CI is not less than the defined non-inferiority limit. The non-inferiority between different vaccine formulations will also be assessed.

#### 16.2.4.2. ANTI-HPV IGG ANTIBODY SEROCONVERSION RATE

The differences in the seroconversion rate at Month 3 and Month 7 will be summarized for each antigen between each HPV9 study group (High, Medium and Low) against Gardasil 9 along with the corresponding 2-sided 95% CI will be reported. The differences in the seroconversion rate at Month 3 and Month 7 between each antigen and HPV9 study group will also be assessed.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx

Author: PPD 3.0 Version Number:


Template No.: CS TP BS016 Revision 7 Reference: CS\_WI\_BS005




# 16.2.4.3. ANTI-HPV NEUTRALIZING ANTIBODY TITERS BETWEEN GROUP ASSESSMENT Anti-HPV neutralizing antibody titers at Month 3 and Month 7 (at least 150 participants in each group) for each antigen.

For each antigen an adjusted GMT and GMT ratio with 2-sided 95% CI for intervention group which is derived from an ANOVA model on log10 transformed titer will be tabulated for anti-HPV neutralizing antibody titer adjusted for country effect. The analysis will be performed at Month 3 and at Month 7, summarised for the prevaccination status of seronegative, seropositive and total. The model will be based on the data from all groups, will include study group and country as a fixed effect and will be based on the PPS. The non-inferiority of different vaccine formulations to the control group will be assessed if the lower limit of the 2-sided 95% CI is not less than the defined non-inferiority limit. The non-inferiority between different vaccine formulations will also be assessed.

### 16.2.4.4. ANTI-HPV NEUTRALIZING ANTIBODY SEROCONVERSION RATE

The differences in the seroconversion rate at Month 3 and Month 7 will be summarized for each antigen between each HPV9 study group (High, Medium and Low) against Gardasil 9 along with the corresponding 2-sided 95% CI will be reported. The differences in the seroconversion rate at Month 3 and Month 7 between each antigen and HPV9 study group will also be assessed.

## 16.2.4.5. COMPARISON OF ANTI-HPV IGG ANTIBODY CONCENTRATION AND ANTI-HPV NEUTRALIZING ANTIBODY TITERS

A qualitative comparison between the ant-HPV IgG antibody concentration and the anti-HPV neutralizing antibody titers will be performed for each antigen by timepoint on all the PPS (except Month 6 and Month 12). This will be performed on each timepoint and antigen where both the anti-HPV IgG antibody concentration and the anti-HPV neutralizing antibody titer will be available. The agreement rate of the 2 results will be summarized and presented along with the kappa and the kappa p-value. The larger the kappa value (close to 1) the better the agreement between the two tests. The McNemar p-value will also be summarized.

## 16.3. Tertiary Immunogenicity

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005






## 16.4. Sensitivity Immunogenicity Variables & Derivations

Sensitivity analysis will be performed on the PPS only.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




The analysis for anti-HPV IgG antibody concentration (section 16.2.3.1), anti-HPV neutralizing antibody titers between group assessment (section 16.2.4.1), anti-HPV neutralizing antibody titers (section 16.2.3.3), anti-HPV neutralizing antibody titers between group assessment (section 16.2.4.3) and the correlation between anti-HPV IgG antibody concentration and anti-HPV neutralizing antibody titers (section ) will all be performed for the sensitivity analysis. The corresponding figures will also be presented for the sensitivity analysis.

The concentration/titer below the assay cut-off will be assigned to half the cut-off for the purpose of GMC/GMT computation. Concentration/titer above the ULOQ will not be imputed. Concentration below the ULOQ for the RCC will not be imputed for the ECL

## 17. SAFETY AND REACTOGENICITY OUTCOMES

## 17.1. Primary Safety and Reactogenicity

## 17.1.1. Primary Safety and Reactogenicity Variables & Derivations

The primary safety and reactogenicity endpoints are:

- Solicited events:
  - Percentage of participants reporting each solicited administration site event assessed as Grade 3 in terms of intensity within 7 days (Day 1 – Day 7) after each vaccine dose
  - Percentage of participants reporting each solicited systemic event assessed as Grade 3 in terms of intensity within 7 days (Day 1 – Day 7) after each vaccine dose
- Unsolicited adverse events:
  - Percentage of participants reporting unsolicited adverse event assessed as Grade 3 in terms of intensity classified by MedDRA within 28 days (Day 1 – Day 28) after each vaccine dose
- Serious adverse events (SAEs):
  - Percentage of participants reporting SAEs classified by MedDRA from first vaccination up to study end
- Safety laboratory parameters (Step 1 participants):
  - Percentage of participants presenting clinically relevant abnormalities in each biochemical and hematological parameter at Day 7 post-dose 1.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## 17.1.2. Intercurrent Event Handling and Data Imputation for Primary Efficacy Variable(s)

See Table A:.

## 17.1.3. Primary Analysis of Primary Safety and Reactogenicity Variables

The primary safety and reactogenicity analysis will be performed for the ES.

#### 17.1.3.1. SOLICITED EVENTS

For each study group and overall and each solicited event, the incidence rate (frequencies and percentages) of vaccinated participants with solicited administration site events (pain at injection site, redness at injection site and swelling at injection site) and systemic events (fever, headache, myalgia, arthralgia and fatigue) assessed as Grade 3 in intensity within 7 days after each vaccine administration will be summarized over the whole vaccination course with the exact 95% CI. The number of solicited events will be summarized at the maximum severity per participant. Each solicited event will be counted once regardless of the number of days the event occurred. The percentages will be out of the number of participants in the ES for each period (after first vaccine dose, after second vaccine dose, after third vaccine dose, overall (dose) and overall (participant)) except the overall dose. The overall dose will be out of the total number of doses in the ES.

Intensity scales for solicited events will be assessed as follows:

| Adverse Event | MedDRA<br>Preferred Term | Intensity<br>Grade | Parameter |
|---|---|---|---|
| | Administration site pain | 1 | Mild: Any pain neither interfering with nor preventing normal everyday activities |
| Pain at Injection Site | (10058049) | 2 | Moderate: Painful when limb is moved and interferes with everyday activities |
| | | 3 | Severe: Significant pain at rest. Prevents normal everyday activities. |
| Redness at Injection | Administration site erythema (10074796) | 1 | Mild: > 0 - ≤ 20 mm |
| Site | | 2 | Moderate: > 20 - ≤ 50 mm |
| | | 3 | Severe: > 50 mm |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| Adverse Event | MedDRA<br>Preferred Term | Intensity<br>Grade | Parameter |
|---|---|---|---|
| Swelling at Injection | Administration site swelling (10075107) | 1 | Mild: > 0 - ≤ 20 mm |
| Site | (100/010/) | 2 | Moderate: > 20 - ≤ 50 mm |
| | | 3 | Severe: > 50 mm |
| | Pyrexia (10037660) | 1 | Mild: ≥ 37.5°C (≥99.5°F) - ≤ 38.0°C (≥100.4°F) |
| Temperature | | 2 | Moderate: > 38.0°C (≥100.4°F) - ≤ 39.0°C (≥102.2°F) |
| | | 3 | Severe: > 39.0°C (≥ 102.2°F) |
| | Headache (10019211) | 1 | Mild: Headache that is easily tolerated |
| Headache | | 2 | Moderate: Headache that interferes with normal activity |
| | | 3 | Severe: Headache that prevents normal activity |
| | Fatigue (10016256) | 1 | Mild: Fatigue that is easily tolerated |
| Fatigue | | 2 | Moderate: Fatigue that interferes with normal activity |
| | | 3 | Severe: Fatigue that prevents normal activity |
| | Arthralgia<br>(10003239) | 1 | Mild: Arthralgia that is easily tolerated |
| Arthralgia | | 2 | Moderate: Arthralgia that interferes with normal activity |
| | | 3 | Severe: Arthralgia that prevents normal activity |
| Make | Myalgia<br>(10028411) | 1 | Mild: Myalgia that is easily tolerated |
| Myalgia | | 2 | Moderate: Myalgia that interferes with normal activity |
| | | 3 | Severe: Myalgia that prevents normal activity |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




#### 17.1.3.2. Unsolicited Events

For each study group and overall, the incidence rates (frequencies and percentages) of participants/events with unsolicited AEs, assessed as Grade 3 and Grade 3 related in intensity assessed by MedDRA occurring within 28-days (Days 1-28) after each vaccine administration will be summarized by SOC and PT over the whole vaccination course with the exact 95% CI. The percentages will be out of the number of participants in the ES for each vaccine dose (after first vaccine dose, after second vaccine dose, after third vaccine dose, overall (dose) and overall (participant)) expect the overall dose. The overall dose will be out of the total number of doses in the ES.

Unsolicited events will be coded using MedDRA central coding dictionary, version 26.0 or higher. Unsolicited events will be described using frequency and percentage.

Unsolicited events will be grouped by SOC and PT and summarized by intervention at time of onset of the event. The summary tables will present the number and percentage of total participants and number of events, by SOC and by PT for each intervention group.

For the summaries of unsolicited events, participants who experience the same AE (in terms of the MedDRA SOC and PT) more than once will only be counted once for that event in the number of participants but all occurrences of the same event will be counted in the number of events.

### 17.1.3.3. SERIOUS ADVERSE EVENTS

For each study group and overall, the incidence rates (frequencies and percentages) of participants/events with SAEs from first vaccination up to Month 12 will be summarized by SOC and PT over the whole vaccination course with the exact 95% CI. The incidence rates (frequencies and percentages) of participants with SAEs causally related to study vaccine, fatal SAEs and causally related fatal SAEs occurring post-dose of study interventions will also be presented. Serious AEs will be recorded on the "Expedited Adverse Events" page of the eCRF.

#### 17.1.3.4. LABORATORY PARAMETERS OUTSIDE NORMAL RANGE

For each study group and overall, the percentage of participants in Step 1 outside the defined normal ranges for each biochemical and hematological parameter measured in the study at Day 7 after the first vaccination will be tabulated with exact 95% CI.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Therefore.


## 17.2. Secondary Safety and Reactogenicity

The secondary safety and reactogenicity analyses will be performed for the ES.

## 17.2.1. Secondary Safety and Reactogenicity Variables & Derivations

The secondary safety and reactogenicity endpoints are:

- Solicited events:
  - Percentage of participants reporting each solicited administration site event within 7 days (Day 1 Day 7) after each vaccine dose
  - Percentage of participants reporting each solicited systemic event within 7 days (Day 1 Day 7) after each vaccine dose
- Unsolicited adverse events:
  - Percentage of participants reporting unsolicited adverse event within 28 days (Day 1 Day 28) after each vaccine dose
- Potential immune-mediated disease (pIMDs)
  - Percentage of participants reporting pIMDs from first vaccination up to study end. A pIMD is an Adverse Event of Special Interest (AESI)
- Pregnancy outcomes
  - Percentage of participants who experienced pregnancy and their outcomes from Day 1 of pregnancy up to study end.

## 17.2.2. Intercurrent Event Handling and Data Imputation for Secondary Safety and Reactogenicity Variable(s)

See Table A:.

## 17.2.3. Analysis of Secondary Safety and Reactogenicity Variables

## 17.2.3.1. SOLICITED EVENTS

For each study group and overall and each solicited event, the incidence rate (frequencies and percentages) of vaccinated participants with solicited administration site events (pain at injection site, redness at injection site and swelling at injection site) and systemic events (fever, headache, myalgia, arthralgia and fatigue) within 7 days after

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




each vaccine administration will be summarized (any, leading to medical advice) over the whole vaccination course with the exact 95% CI. The completeness defined as the percentage of vaccinated participants who documented presence/absence of each event as well as the daily prevalence of each symptom among vaccinated participants who documented presence /absence of the event on that day will be provided. The percentages will be out of the number of participants who have at least one documented event (either present or absent). The number of solicited events will be summarized at the maximum severity per participant. Each solicited event will be counted once regardless of the number of days the event occurred. The number of solicited events will also be summarized by severity. The percentages will be out of the number of participants in the ES for each period (after first vaccine dose, after second vaccine dose, after third vaccine dose, overall (dose) and overall (participant)) expect the overall dose. The overall dose will be out of the total number of doses in the ES.

The duration of each Grade 3 solicited event (split between solicited administration events and systemic events) will be summarized. The duration of the event is defined as the number of days that a participant had an event, for example if an event occurs on day 2 and 4 but the event did not occur on day 3 (or was not captured in the eDiary) then the duration is considered as 2 days. The duration will be summarized numerically (with n, mean, STD, median, minimum and maximum) and also the frequency (the number of events that had a duration of 1, 2, 3,4, >=5 days).

#### 17.2.3.2. Unsolicited Events

For each study group and overall, the incidence rates (frequencies and percentages) of participants/events with unsolicited AEs (any, related, leading to medical attention), occurring within 28-days (Days 1-28) after each vaccine administration and overall will be summarized by SOC and PT with the exact 95% CI. The number of unsolicited events will also be summarized by severity. The percentages will be out of the number of participants in the ES for each period (after first vaccine dose, after second vaccine dose, after third vaccine dose, overall (dose) and overall (participant)) expect the overall dose. The overall dose will be out of the total number of doses in the ES.

Causality, as indicated by the Investigator is classed as "related" and "not related" to HPV vaccine. A "related" AE is defined as an AE with a relationship to study intervention as "related". If a participant reports the same AE more than once within that SOC/PT, the AE with the worst-case relationship to study intervention will be used in the corresponding relationship summaries for each vaccination group.

Unsolicited events will be coded using MedDRA central coding dictionary, version 26.0 or higher. Unsolicited events will be described using frequency and percentage.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




Unsolicited events will be grouped by SOC and PT and summarized by intervention at time of onset of the event. The summary tables will present the number and percentage of total participants and number of events, by SOC and by PT for each intervention group.

For the summaries of unsolicited events, participants who experience the same AE (in terms of the MedDRA SOC and PT) more than once will only be counted once for that event in the number of participants but all occurrences of the same event will be counted in the number of events.

#### 17.2.3.3. POTENTIAL IMMUNE-MEDIATED DISEASE

For each study group and overall, the incidence rates (frequencies and percentages) of participants/events with pIMDs and pIMDs causally related to study vaccine from first vaccination up to study end will be summarized (any and related) over the whole vaccination course with the exact 95% CI.

#### 17.2.3.4. PREGNANCY

For each study group and overall, the percentage of participants who experienced pregnancy during the entire study and around each vaccination (30 days before and 45 days after each vaccination) will be summarized along with their outcomes.

## 17.3. Laboratory Parameters

Scheduled clinical safety laboratory parameters will be summarized at each visit by grade (grade 0, 1, 2, 3 and 4) according to Table 13 of the protocol. These include:

- Hematology: hemoglobin, hemoglobin change from baseline, White Blood Cell (WBC) increase, WBC decrease, lymphocyte decrease, neutrophils decrease, eosinophils and platelet decrease
- Chemistry: Blood Urea Nitrogen (BUN), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT)

Box plots of the above summary will be presented for the iSRC analysis.

## 18. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




- Physical examination
- Vital signs
- Body temperature

These domains and/or variables will not be summarized or presented, but will be available in the clinical study database, SDTM and/or ADaM datasets. Vital signs and body temperature will be presented in a listing.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




## 19. REFERENCES

Clopper CJ, Pearson ES. The use of confidential or fiducial limits illustrated in the case of the binomial. Biometrika 1934; 26:404-413

Nauta J. Statistics in Clinical Vaccine Trials. 2010. Heidelberg: Springer.

Brown et all. Concordance assessment between a multiplexed competitive Luminex immunoassay, a multiplexed IgG Luminex immunoassay, and a pseudovirion-based neutralization assay for detection of human papillomaviruse types 16 and 18. 2014.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

## **IQVIA Output Conventions**

Outputs will be presented according to the following IQVIA Output Conventions

**Document Headers** 

All TFL is to include the following header:

GSK Vaccines Vaccine: HPV

Study 213749 (HPV9) - DELIVERY DESIGNATION

where delivery designation is the name of the current delivery, e.g., DRY-RUN, FINAL ANALYSIS REPORT, etc

## **Dates & Times**

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

## **Spelling Format**

English US

## **Presentation of Treatment Groups**

For outputs, treatment groups will be represented as follows and in the given order:

| Treatment Group | For Tables and Figures | For Listings (include if different to tables) |
|---|---|---|
| HPV9High | HPV9 High | HPV9 High |

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| Treatment Group | For Tables and Figures | For Listings (include if different to tables) |
|---|---|---|
| HPV9Med | HPV9 Med | HPV9 Medium |
| HPV9Low | HPV9 Low | HPV Low |
| Gar9 | Gardasil 9 | Gardasil 9 |

## **Presentation of Visits**

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Visit 1 (Day 1) | Day 1 |
| Visit 2 (Day 7) | Day 7 |
| Visit 3 (Month 2) | Month 2 |
| Visit 4 (Month 3) | Month 3 |
| Visit 5 (Month 6) | Month 6 |
| Visit 6 (Month 7) | Month 7 |
| Visit 7 (Month 12) | Month 12 |

## Listings

All listings will be ordered by the following (unless otherwise indicated in the template):

- Randomized treatment group (or treatment received if it's a safety output), first by HPV9High then HPV9Med, then HPV9Low and then Gardasil9
- Center-subject ID,
- Date (where applicable),

•

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


### **DECIMAL PLACES**

Decimal places for categorical data

- For percentages one decimal will be displayed
- Differences in percentages and their corresponding confidence limits will be displayed with one more
  decimal than the maximum number used to display the individual percentages, for example the
  difference between two percentages displayed with one decimal will be displayed with two decimals.

Decimal places for Demographic and baseline characteristics will be as follows:

The mean, median, and SD for continuous baseline characteristics (age) will be presented with one decimal.

Serological Summary Statistics

The number of decimals used when displaying geometric mean concentrations (GMC) and their confidence limits is shown in the following table:

| GMC value | Number of decimals |
|----------------|--------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMC values of <0.1 appear in the same table as values of >=0.1 and <10 3 decimals should be displayed for both.

GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

Document: \quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## APPENDIX 2. PARTIAL DATE CONVENTIONS

Imputed dates will NOT be presented in the listings.

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30th.

The following exceptions apply:

- Adverse event start dates with missing day:
  - o If the event starts in the same month as the study intervention, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the study intervention given during that month.
- Adverse event start dates with missing day and month:
  - o If the event starts in the same year as study intervention, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the study intervention given during that year. If 'before vaccination' is selected, the imputed date will be one day before the) study intervention given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## **Algorithm for Prior / Concomitant Medications:**

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= study med end date, assign as concomitant |

Document: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= study med end date, assign as concomitant |
| | Missing | If stop date is missing could never be assumed a prior medication If start date <= study med end date, assign as concomitant |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= study med end date, assign as concomitant |
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= study med end date, assign as concomitant |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date is missing could never be assumed a prior medication If start date <= study med end date, assign as concomitant |
| Missing | Known | If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK\_213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day |
| | | unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date, assign as concomitant |
| | Missing | Assign as concomitant |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Documentation\SAP\GSK 213749(HPV9-AS04-

001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

## TABLE, FIGURES AND LISTINGS SHELLS

## 213749 (HPV9-AS04-001)

A Phase 1/2 randomized, observer-blinded, multi-country study to evaluate safety and immunogenicity of investigational adjuvanted human papillomavirus vaccine in females (16 to 26 years of age)

AUTHOR:

VERSION NUMBER AND DATE: V3.0, 05FEB2024

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0

Author: Version Date: 05FEB2024

## TABLE, LISTINGS AND FIGURES SHELLS SIGNATURE PAGE

Table, listing and Figures Shells V3.0 (Dated 05FEB2024) for Protocol 213749 (HPV9-AS04-001)

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|-------------------------------|---------------|------------------|
| Author: | PPD | Refer to ePPD | uary 6, 2024 |
| Position: | Associate Director Biostatist | ics | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|--------------|------------------------|-----------|------------------|
| Approved By: | PPD | PPD | bruary 8, 2024 |
| Position: | Senior Biostatistician | | |
| Company: | IQVIA | | |
| Approved By: | PPD | PPD | February 5, 202 |
| Position: | Project Statistician | | |
| Company: | GSK | | |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number:

3.0

Author:

## MODIFICATION HISTORY

| Unique Identifier for this Version 1.0 | Date of the Document Version 03AUG2022 | Author PPD | Significant Changes from Previous Authorized Version Not Applicable – First Version |
|---|---|---|---|
| 2.0 | 21JUL2023 | PPD | Updates based on Statistical Analysis Plan V2.0. Including list of outputs required for the interim analysis and the headline results |
| 3.0 | 05FEB2024 | PPD | Updates following the first interim analysis. New outputs – demography tables for each of the Per Protocol Sets, concordance analysis table and duration of grade 3 solicited events tables |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\
GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx
PPD \\quad \text{Varsion Number:}

3.0 Version Number:

Author:

| List of Outputs Required for Interim Analysis7 |
|---|
| Table 14.1.1.1: Summary of Participant Disposition (Enrolled Set) |
| Table 14.1.1.2: Number of Participants at each visit (Exposed Set) |
| Table 14.1.1.3: Number and Percentage of Participants Discontinued due to COVID-19 (Exposed Set) |
| Table 14.1.1.4: Number of Participants Enrolled by Age Category (Exposed Set) |
| Table 14.1.2: Summary of Protocol Deviations Leading to Elimination from Per Protocol Set (Exposed Set) |
| Table 14.1.3: Summary of Analysis Sets (Enrolled Set) |
| Table 14.1.4.1.1: Summary of Demographic and Baseline Characteristics (Exposed Set) |
| Table 14.1.4.1.2: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Day 1) |
| Table 14.1.4.1.3: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 2) |
| Table 14.1.4.1.4: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 3)20 |
| Table 14.1.4.1.5: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 6) |
| Table 14.1.4.1.6: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 7) |
| Table 14.1.4.1.6: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 1) |
| Table 14.1.4.2: Summary of Medical History (Exposed Set) |
| Table 14.1.4.3: Summary of Concomitant Vaccinations (Exposed Set) |
| overall (Exposed Set) |
| Table 14.1.5: Study Vaccine Administration (Exposed Set) |
| Table 14.1.6: Summary of Important Protocol Deviations Leading to Elimination from any analyses (Enrolled Set)27 |
| Table 14.2.1.1: Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, |
| Month 6, Month 7 and Month 12 (Per Protocol Set) |
| Table 14.2.1.2: Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, |
| Month 6, Month 7 and Month 12 (Exposed Set) |
| Table 14.2.2.1.1: Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between Groups (HPV group |
| [different potencies - Low, Med, High] divided by Gardasil 9 group) (Per Protocol Set) |
| Table 14.2.2.1.2: Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between HPV Groups (Per |
| Protocol Set) |
| Table 14.2.2.2: Differences of anti-HPV IgG Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 |
| between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group) (Per Protocol Set) |
| Table 14.2.2.3: Summary of anti-HPV Neutralizing Antibody GMTs and seropositivity for each antigen at Day 1, Month 2, |
| Month 3 and Month 7 (Per Protocol Set) |
| Table 14.2.2.4.1: Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between Groups |
| (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group) (Per Protocol Set) |
| Table 14.2.2.4.2: Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between HPV |
| Groups (Per Protocol Set) |
| Table 14.2.2.5: Differences of anti-HPV Neutralizing Antibody Seroconversion Rate for each antigen at Month 3 and Month |
| 7 between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group) (Per Protocol Set)43 |
| Table 14.2.2.6: Correlation between anti-HPV Immunoglobulin Antibody Concentration and anti-HPV Neutralizing Antibody |
| Titers for each antigen at Day 1, Month 2, Month 3 and Month 7 (Per Protocol Set) |
| Table 14.2.2.7: Functional Relationship between the Assay Methods for each antigen (Per Protocol Set) |
| Table 14.2.2.8 Summary of qualitative comparison between anti-HPV Immunoglobulin Antibody Concentration and anti-HPV |
| Neutralizing Antibody Titers for each antigen by time point analysis (Per Protocol Set) |
| \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


05FEB2024

3.0

CCI

```
Table 14.3.1.1: Overall Summary of Grade 3 Solicited Administration Site Events and Solicited Systemic Events Reported
Table 14.3.1.2.1: Number and Percentage of Participants of each Grade 3 Solicited Administration Site Events Reported
Table 14.3.1.2.2: Summary of duration of Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7)
Table 14.3.1.2.3: Number and percentage of participants with Grade 3 Solicited Administration Site Events Reported
Table 14.3.1.3.1: Number and Percentage of Participants of each Grade 3 Solicited Systemic Events Reported within 7
Table 14.3.1.3.2: Summary of duration of Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each
Table 14.3.1.3.3: Number and percentage of participants with Grade 3 Solicited Systemic Events Reported within 7 days
Table 14.3.1.4: Summary of Participants with any Grade 3 Unsolicited Events and Serious Adverse Events (Exposed Set) .67
Table 14.3.1.5: Number and Percentage of Participants of each Grade 3 Unsolicited Adverse Events Reported within 28
days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set) ..........69
Table 14.3.1.6: Number and Percentage of Participants of causally related Grade 3 Unsolicited Adverse Events Reported
within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set) 71
Table 14.3.1.7: Number and Percentage of Participants of Serious Adverse Events Reported up to Study End by System
Table 14.3.1.8: Number and Percentage of Participants of causally related Serious Adverse Events Reported up to Study
Table 14.3.1.9: Number and Percentage of Participants of fatal Serious Adverse Events Reported up to Study End by
Table 14.3.1.10: Number and Percentage of Participants of causally related fatal Serious Adverse Events Reported up to
Table 14.3.1.11: Number and Percentage of Participants of Laboratory Parameters Outside normal range at Day 7 after the
Table 14.3.2.1: Overall Summary of Solicited Administration Site Events and Solicited Systemic Events Reported within 7
Table 14.3.2.2: Number and Percentage of Participants of Solicited Administration Site Events Reported within 7 days
Table 14.3.2.3: Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7)
Table 14.3.2.4: Number and Percentage of Participants of Solicited Administration Site Events Reported within 7 days
Table 14.3.2.5: Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7)
```

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx

Author: Version Number: 3.0

| Table 14.3.2.6.1: Solicited Events, Completeness Analysis, by Administration Site and Systemic Category by Intervention Group and overall (Exposed Set) |
|---|
| (Exposed Set) |
| (Exposed Set) |
| 28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set) |
| Table 14.3.2.7.4: Number and Percentage of Participants with Unsolicited Adverse Events Leading to Medical Attention Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term |
| (Exposed Set) |
| by System Organ Class and Preferred Term (Exposed Set) |
| Table 14.3.2.9.1: Number and Percentage of Participants of Pregnancies Reported up to Study End (Exposed Set)115 Table 14.3.2.9.2: Number and Percentage of Participants of Pregnancies Reported around each Vaccination (Exposed Set) |
| Table 14.3.2.9.3: Number and Percentage of Participants of Pregnancies Outcomes Reported up to Study End (Exposed Set) |
| Table 14.3.3.1: Summary of Laboratory Parameters Grades: Hematology by study group and overall (Exposed Set) |
| Month 2, Month 3, Month 7 and Month 12 (Per Protocol Set) |
| concentrations for each antigen (Per Protocol Set) |
| Listing 16.2.1.2: Participants with Early Withdrawal or Discontinuation due to COVID-19 (Enrolled Set) |
| Listing 16.2.1.4: Inclusion and Exclusion Criteria at Enrolment (Enrolled Set) |
| Listing 16.2.4.1: Demographics and Other Baseline Characteristics (Enrolled Set) |
| Listing 16.2.4.3: Prior and Concomitant Vaccinations (Enrolled Set) |
| Listing 16.2.5: Vaccine Administration (Enrolled Set) |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\
GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

\text{Version Number:}

Author:


05FEB2024 Version Date:

3.0

## GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

| Listing | 16.2.6.2: | Listing of anti-HPV IgG Neutralizing Antibody Titers for each Participant (Enrolled Set) | . 139 |
|---|---|---|---|
| Listing | 16.2.7.1: | Solicited Administration Site Events (Enrolled Set) | . 140 |
| Listing | 16.2.7.2: | Solicited Systemic Events (Enrolled Set) | . 142 |
| | | Unsolicited Adverse Events (Enrolled Set) | |
| Listing | 16.2.7.4: | Unsolicited Adverse Events Leading to Withdrawal or Discontinuation from Study (Enrolled Set) | . 144 |
| Listing | 16.2.7.5: | Serious Adverse Events (Enrolled Set) | . 145 |
| Listing | 16.2.7.6: | All Serious Adverse Events Leading to Withdrawal or Discontinuation from Study (Enrolled Set) | .14 |
| Listing | 16.2.7.7: | Potential Immune-Mediated Disease Events (Enrolled Set) | .14 |
| | | Laboratory Results (Enrolled Set) | |
| Listing | 16.2.8.2: | Pregnancies - Follow up Report (Enrolled Set) | . 149 |
| Listing | 16.2.8.3: | Vital Signs (Enrolled Set) | . 153 |
| _ | | Body Temperature (Enrolled Set) | |

## List of Outputs Required for Interim Analysis

The below file contains the ToC of the outputs that are required for the iSAC, and whether they are synopsis tables or intext tables. It also displays which outputs will also be created separately for the sensitivity analysis.



\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author: Version Date: 05FEB2024

## Table 14.1.1.1: Summary of Participant Disposition (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.1.1
Summary of Participant Disposition
Enrolled Set

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| | 40.1 | , , | , , | , | , | , , |
| Number of participants enrolled | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants enrolled but not vaccinated | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants vaccinated | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Participants who completed the study | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Participants who discontinued the study | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Reason for discontinuing the study | | | | | | |
| Adverse event requiring expedited reporting | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Pregnancy | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Unsolicited AE | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Solicited AE | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Withdrawal by participant | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Migrated/moved from the study area | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Lost to follow up | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Study termination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Withdrew due to COVID-19 pandemic | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Other | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. AE = Adverse Event. COVID-19 = Coronavirus Disease 2019.

N is the number of participants in the Enrolled Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

A participant is considered to have completed the study if he/she returns for the last visit/contact or is available for the last scheduled procedure/contact as described in the protocol

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.1.1.1 Summary of Participant Disposition Enrolled Set

| HPV: | HPV9 Medium | HPV9 High |
|------|-------------|-----------|
| (N= | (N=XXX) | (N=XXX) |

Programming Notes

Output ID: DS0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\_213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.1.1.2: Number of Participants at each visit (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.1.2

Number of Participants at each visit

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Participants attending each | visit: | | | | | |
| Visit 1 (Day 1) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 2 (Day 7)* | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 3 (Month 2) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 4 (Month 3) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 5 (Month 6) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 6 (Month 7) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 7 (Month 12) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

\* = Step 1 participants only

Programming Notes

Output ID: DS0002

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.1.1.3: Number and Percentage of Participants Discontinued due to COVID-19 (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.1.3

Number and Percentage of Participants Discontinued due to COVID-19

Exposed Set

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Participants discontinued/withdrew from the study due to | | | | | | |
| COVID-19 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Participants missed visit due to COVID-19 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 1 (Day 1) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 2 (Day 7)* | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 3 (Month 2) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 4 (Month 3) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 5 (Month 6) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 6 (Month 7) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 7 (Month 12) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. COVID-19 = Coronavirus disease 2019.

N is the number of participants in the Exposed Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

\* = Step 1 participants only

Programming Notes

Output ID: DS0003

 $[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749]$ 

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.1.1.4: Number of Participants Enrolled by Age Category (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| Characteristic | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Age category | | | | | | |
| Preterm newborn - gestational age < 37 weeks | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Newborn (0-27 days) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Infant and toddlers (28 days to 23 months) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Children (2-11 years) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Adolescents (12-17 years) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| From 18 - 64 years | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| From 65 - 84 years | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Over 85 years | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Enrolled Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Programming Notes

Output ID: DS0004

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.1.2: Summary of Protocol Deviations Leading to Elimination from Per Protocol Set (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.2 Summary of Protocol Deviations Leading to Elimination from Per Protocol Set Exposed Set

| | | HPV9<br>High | HPV9<br>Medium | HPV9<br>Low | Gardasil<br>9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX |
| Withdrawals at Day 1 | n<br>(%) | | | | | |
| withdiawais at bay i | | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| AE requiring expedited reporting | n | | | | | |
| im rodurring onboaroom robororing | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Pregnancy | n | , , | , , | , , | | , , |
| -31 | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Unsolicited AE (non-serious) | n | | , , | , , | , , | , , |
| · | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Solicited AE | n | () | () | () | () | () |
| | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Not willing to be vaccinated | n<br>(%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | (%)<br>n | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Discontinued study treatment due to COVID-19 pandemic | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n ( ° ) | A (A.A) | Α (Δ.Δ) | Α (Δ•Α) | Δ (Δ•Δ) | Δ (Δ.Δ) |
| Other | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | . , | , , | , , | , , | | , , |
| | n | | | | | |
| Eliminations at Day 1 | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n | , , | , | , | , , | , , |
| Informed consent criteria | (응) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| To all was to an another of a | n | | | | | |
| Inclusion criteria | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Exclusion criteria | n | | | | | |
| EXCLUSION CITCELLA | (응) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Concomitant medication | n | | | | | |
| CONCOMITERITE MENTERALION | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.1.2 Summary of Protocol Deviations Leading to Elimination from Per Protocol Set Exposed Set

| Laboratory assessment | n<br>(%) | High<br>(N=XXX) | Medium (N=XXX) | Low | 9 | Total<br>(N=XXX |
|---|---|---|---|---|---|---|
| • | | (N=XXX) | (N=XXX) | (N=XXX) | / NT 3/3/3/ | |
| • | | | | | (N=XXX) | ) |
| • | | | | | | |
| | | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Study procedure | n | | | | | |
| study procedure | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Safety | n | | | | | |
| 1 | (용) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Randomization | n<br>(%) | v (v v) | v (v v) | v (v v) | v (v v) | v (v ··· |
| | (%)<br>n | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit schedule | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n | A (A•A) | A (A.A) | A (A.A) | A (A.A) | A (A.A) |
| IP conditions | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| ID managed in | n | | | | | |
| IP preparation | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| IP administration | n | | | | | |
| ir daministration | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Subject IP compliance | n | | | | | |
| | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Efficacy | n | ( | ( | ( | ( | |
| - | (응)<br>n | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Subject discontinuation | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n (°) | A (A•A) | A (A.A) | A (A.A) | A (A.A) | A (A.A) |
| Blinding | (응) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n | , , | , , | , , | , , | , |
| Patient Reported Outcomes | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x |
| Other | n | | | | | |
| ocher | (왕) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| mber of participants included in the Per Protocol Set at | n | | | | | |
| y 1 | (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set.

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### 

| HPV9 | HPV9 | HPV9 | Gardasil | Total |
|---------|---------|---------|----------|--------|
| High | Medium | Low | 9 | (N=XXX |
| (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Participants with both a withdrawal and an elimination at the timepoint are summarized in the withdrawals only

Programming Notes

Continue for the following visits: Month 2, Month 3, Month 7 and Month 12 Only present categories which do occur.

Output ID: PD0001

Author:

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

PPD Version Number: 3.0

## Table 14.1.3: Summary of Analysis Sets (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.3
Summary of Analysis Sets
Enrolled Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of participants in enrolled set | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in exposed set | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in per protocol set at day 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in per protocol set at month 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in per protocol set at month 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in per protocol set at month 7 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in <a href="per protoc">per protoc</a> ol set at month 12 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number of participants in CCI | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Enrolled Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Programming Notes

Output ID: AS0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

### Table 14.1.4.1.1: Summary of Demographic and Baseline Characteristics (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| Characteristic | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Age (years) at time of first vaccination | n | х | x | х | x | х<br>х.х |
| | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | (x.xx) |
| | Median | X • X | X . X | X . X | X • X | X.X |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Age category (years | | | | | | |
| <18 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=18 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Race | | | | | | |
| Black or African American | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| American Indian or Alaska Native | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Asian | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Native Hawaiian or other Pacific Islander | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| White | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Other* | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Missing | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Ethnicity | | | | | | |
| Hispanic or Latino | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Not Hispanic nor Latino | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


# $\begin{array}{c} \text{Table 14.1.4.1.1} \\ \text{Summary of Demographic and Baseline Characteristics} \\ \text{Exposed Set} \end{array}$

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| Characteristic | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

 $\ensuremath{\text{n}}$  is the number of participants in each category.

Percentages are calculated as  $100 \times n/N$ .

\* Other includes participants with multiple race categories.

Programming Notes

Missing row only included if 1 or more participant have missing information

Output ID: DM0001

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


Version Date: 05FFB2024

## Table 14.1.4.1.2: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Day 1)

Table 14.1.4.1.2

Summary of Demographic and Baseline Characteristics

Per Protocol Set at Day 1

DM0002: This output uses shell DM0001 [Table 14.1.4.1.1]

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Per Protocol Set at Day 1.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

\* Other includes participants with multiple race categories.

 ${\it Programming Notes}$ 

• Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information

## Table 14.1.4.1.3: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 2)

Table 14.1.4.1.3

Summary of Demographic and Baseline Characteristics

Per Protocol Set at Month 2

DM0002: This output uses shell DM0001 [Table 14.1.4.1.1]

Source: Listing xx.x.x.x Abbreviations: HPV = Human Papillomavirus. N is the number of participants in the Per Protocol Set at Month 2. n is the number of participants in each category. Percentages are calculated as  $100 \, * \, n/N$ . \* Other includes participants with multiple race categories.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Programming Notes

• Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information

### Table 14.1.4.1.4: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 3)

Table 14.1.4.1.4

Summary of Demographic and Baseline Characteristics
Per Protocol Set at Month 3

DM0002: This output uses shell DM0001 [Table 14.1.4.1.1]

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Per Protocol Set at Month  $3. \,$ 

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

\* Other includes participants with multiple race categories.

Programming Notes

• Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information

### Table 14.1.4.1.5: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 6)

Table 14.1.4.1.5

Summary of Demographic and Baseline Characteristics

Per Protocol Set at Month 6

DM0002: This output uses shell DM0001 [Table 14.1.4.1.1]

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Version Date:

05FFB2024

Source: Listing xx.x.x.x Abbreviations: HPV = Human Papillomavirus. N is the number of participants in the Per Protocol Set at Month 6. n is the number of participants in each category. Percentages are calculated as 100 \* n/N. \* Other includes participants with multiple race categories. Programming Notes · Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information Table 14.1.4.1.6: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 7) Table 14.1.4.1.6 Summary of Demographic and Baseline Characteristics Per Protocol Set at Month 7 DM0002: This output uses shell DM0001 [Table 14.1.4.1.1] Source: Listing xx.x.x.x Abbreviations: HPV = Human Papillomavirus. N is the number of participants in the Per Protocol Set at Month 7. n is the number of participants in each category. Percentages are calculated as 100 \* n/N. \* Other includes participants with multiple race categories. Programming Notes · Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information Table 14.1.4.1.7: Summary of Demographic and Baseline Characteristics (Per Protocol Set at Month 12) \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx Version Number: 3.0

Author:

# Table 14.1.4.1.7 Summary of Demographic and Baseline Characteristics Per Protocol Set at Month 12

DM0002: This output uses shell DM0001 [Table 14.1.4.1.1]

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Per Protocol Set at Month 12.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

\* Other includes participants with multiple race categories.

#### Programming Notes

Author:

• Replace footnotes in original shell with those listed above Missing row only included if 1 or more participant have missing information


### Table 14.1.4.2: Summary of Medical History (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.4.2
Summary of Medical History
Enrolled Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Participants with medical/vaccination history | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| System Organ Class 1 | | | | | | |
| Preferred term 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Preferred term 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Preferred term 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| System Organ Class 2 | | | | | | |
| Preferred term 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Preferred term 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. Medical history coded using MedDRA version xx.x N is the number of participants in the Enrolled Set. n is the number of participants in each category. Percentages are calculated as 100 \* n/N.

Programming Notes

Output ID: MH0001

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Table 14.1.4.3: Summary of Concomitant Vaccinations (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

# Table 14.1.4.3 Summary of Concomitant Vaccinations Exposed Set

| | HPV9 High | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | n (%)<br>n (%)<br>n (%) | n (%) x (x.x) n (%) x (x.x) n (%) x (x.x) n (%) x (x.x) n (%) x (x.x) | (N=XXX) (N=XXX) n (%) x (x.x) x (x.x) n (%) x (x.x) x (x.x) n (%) x (x.x) x (x.x) n (%) x (x.x) x (x.x) | (N=XXX) (N=XXX) (N=XXX) n (%) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) | (N=XXX) (N=XXX) (N=XXX) (N=XXX) n (%) x (x.x) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) x (x.x) n (%) x (x.x) x (x.x) x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. ATC = Anatomical therapeutic chemical.

N is the number of participants in the Exposed Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Concomitant vaccinations coded using WHO drug dictionary version x.x.

Concomitant vaccinations are any vaccines that the participant received at the time of enrolment or received during the study.

Programming Notes

Output ID: CM0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


## Table 14.1.4.4: Summary of Participants starting a Concomitant Medication within 30 days following each dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### 

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Any medications | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| any antipyretic | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Non prophylastic antinumetic | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Any prophylactic antipyretic | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| North and Alled and a | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Any antibiotic | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


Author:

Version Nate: 05FEB2024

### Table 14.1.5: Study Vaccine Administration (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.1.5 Study Vaccine Exposure Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Exactly 1 dose | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Exactly 2 doses | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Exactly 3 doses | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least 1 dose | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least 2 doses | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set.

n is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Exactly x dose(s) categories are mutually exclusive.

Programming Notes

Output ID: EX0001

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author: Version Date: 05FFB2024

## Table 14.1.6: Summary of Important Protocol Deviations Leading to Elimination from any analyses (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| Category<br>Sub category | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one important protocol deviation | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <each category=""></each> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <each category="" sub=""></each> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the enrolled set.

 $\ensuremath{\text{n}}$  is the number of participants in each category.

Percentages are calculated as 100 \* n/N.

Programming Notes

Output ID: AS0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


Table 14.2.1.1: Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, Month 6, Month 7 and Month 12 (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.1.1

Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, Month 6, Month 7 and Month 12

Per Protocol Set

| | Pre- | | | | | |
|---|---|---|---|---|---|---|
| isit / | vaccination<br>status | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 |
| ay 1 | Seronegative | N | XXX | XXX | XXX | XXX |
| _ | - | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMC (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X.X | X.X | X . X | X.X |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMC | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | Seropositive | N | XXX | XXX | xxx | xxx |
| | - | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMC (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | x.x | x.x | x.x | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMC | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | N | XXX | XXX | xxx | xxx |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMC (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | x.x | X.X | x.x | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMC | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


Version Date: 05FEB2024

3.0

#### Table 14.2.1.1

Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, Month 6, Month 7 and Month 12

Per Protocol Set

| /isit | Pre-<br>vaccination<br>status | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 |
|---|---|---|---|---|---|---|
| | | | 9 | | | |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| onth 2 | Seronegative | N | х | X | x | X |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMC (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X.X | X . X | X . X | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMC | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ltc. | | | | | | |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMC = Geometric Mean Concentration. GSD = Geometric Standard Deviation. LLOQ = Lower Limit of Quantification. ULOQ = Upper Limit of Quantification.

 ${\tt N}$  = number of participants in the Per Protocol Set at each visit and pre-vaccination status.

n (%) = number/percentage of participants with concentration equal or above LLOQ.

95% CI GMC = 95% confidence interval derived using the log10-transformed antibody concentration.

Seronegative is defined as the situation where antibodies are not elevated (i.e, concentrations less than the LLOQ) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOQ) in the serum of participants.

The concentration below the LLOQ will be replaced by half the LLOQ (LLOQ/2). Concentration above the ULOQ will be replaced by the ULOQ.

Programming Notes

Output ID: IM0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.2.1.2: Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, Month 6, Month 7 and Month 12 (Exposed Set)

#### Table 14.2.1.2

Summary of anti-HPV IgG Antibody GMCs and seropositivity for each antigen at Day 1, Month 2, Month 3, Month 6, Month 7 and Month 12 Exposed Set

IM0002: This output uses shell IM0001 [Table 14.2.1.1]

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMC = Geometric Mean Concentration. GSD = Geometric Standard Deviation.

LLOQ = Lower Limit of Quantification. ULOQ = Upper Limit of Quantification.

N = number of participants in the Exposed Set at each visit and pre-vaccination status. n (%) = number/percentage of participants with concentration equal or above LLOQ.

95% CI = 95% confidence interval derived using the log10-transformed antibody concentration.

Seronegative is defined as the situation where antibodies are not elevated (i.e, concentrations less than the LLOO) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOO) in the serum of participants.

The concentration below the assay LLOQ will be replaced by half the LLOQ (LLOQ/2). Concentration above the ULOQ will be replaced by the ULOQ.

#### Programming Notes

- · Replace footnotes in original shell with those listed above
- Table is only required when >5% of participants have been excluded from the PPS when compared with the ES

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells\_V3.0\_05FEB2024.docx


Table 14.2.2.1.1: Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group) (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.1.1

Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group)

Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| Pre-vaccination | | HE | PV9 Group | Garda | asil 9 Group | Group GMC Ratio | |
|---|---|---|---|---|---|---|---|
| status | | N A | Adjusted GMC | N A | Adjusted GMC | Value | 95% CI |
| Seronegative | anti-HPV IgG concentration at Month 3 | | | | | | |
| , | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| Seropositive | anti-HPV IgG concentration at Month 3 | | | | | | |
| - | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | xx.x | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| Total | anti-HPV IgG concentration at Month 3 | | | | | | |
| | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | xx.x | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| Seronegative | anti-HPV IgG concentration at Month 7 | | | | | | |
| - | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |

•••

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


#### Table 14.2.2.1.1

Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group)

Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| Pre-vaccination | HPV9 Group | Gardasil 9 Group | Group GMC Ratio |
|-----------------|----------------|------------------|-----------------|
| status | N Adjusted GMC | N Adjusted GMC | Value 95% CI |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMC = Geometric Mean Concentration.

N = Number of participants with available results

The analysis is based on ANOVA model with log10 transformed anti-gE antibody concentration values as response variable and the study group and country as fixed effects.

Seronegative is defined as the situation where antibodies are not elevated (i.e, concentrations less than the LLOQ) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOQ) in the serum of participants.

95% CI GMC = 95% confidence interval derived using the log-transformed antibody concentration.

The concentration below the assay cut-off will be replaced by half the cut-off (LLOQ/2). Concentration above the ULOQ will be replaced by the ULOQ

Programming Notes

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Output ID: IM0003

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\\ GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells \(\forall V3.0 \) 05FEB2024.docx


## Table 14.2.2.1.2: Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between HPV Groups (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.2.2.1.2 Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between HPV Groups Per Protocol Set

| Pre-<br>vaccination | | First Group | | First Group | | Second Group | | Group GMC Ratio |
|---|---|---|---|---|---|---|---|---|
| status | | N | Adjusted GMC | N A | Adjusted GMC | Value | 95% | CI |
| Seronegative | anti-HPV IgG concentration at Month 3 | | | | | | | |
| beronegaerve | HPV9 High / HPV9 Medium | ХХ | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| Seropositive | anti-HPV IgG concentration at Month 3 | | | | | | | |
| - | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | xx.x | xx.x; | XX. |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX. |
| Total | anti-HPV IgG concentration at Month 3 | | | | | | | |
| | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |
| Seronegative | anti-HPV IgG concentration at Month 7 | | | | | | | |
| - | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | xx.x | xx.x; | XX.X |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | xx.x | xx.x; | XX.X |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; | XX.X |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0


3.0

#### Table 14.2.2.1.2

Ratio of anti-HPV IgG Antibody GMCs for each antigen at Month 3 and Month 7 between HPV Groups

Per Protocol Set

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMC = Geometric Mean Concentration.

N = Number of participants with available results

The analysis is based on ANOVA model with log10 transformed anti-gE antibody concentration values effect as response variable and the study group and country as fixed effects.

Seronegative is defined as the situation where antibodies are not elevated (i.e, concentrations less than the LLOQ) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOQ) in the serum of participants.

95% CI = 95% confidence interval derived using the log-transformed antibody concentration.

The concentration below the assay cut-off will be replaced by half the cut-off (LLOQ/2). Concentration above the ULOQ will be replaced by the ULOQ

Programming Notes

Programming Notes

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Output ID: IM0003

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:

Version Pate: 05FEB2024

Table 14.2.2.2: Differences of anti-HPV IgG Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group) (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.2

Differences of anti-HPV IgG Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - [Low, Med, High] and Gardasil9 group]

Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| | First | t Stud | ly Group | Secon | d Sti | ıdy Group | Di | fferen | ce |
|---|---|---|---|---|---|---|---|---|---|
| | N | n | (%) | N | r | ૧ (%) | % | 95% | CI |
| Seroconversion Rate at Month 3 | | | | | | | | | |
| HPV9 High - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 Medium - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 Low - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 High - HPV9 Low | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | XX.X; | XX.X |
| HPV9 Medium - HPV9 Low | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 High - HPV9 Medium | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | XX.X; | XX.X |
| Seroconversion Rate at Month 7 | | | | | | | | | |
| HPV9 High - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 Medium - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 Low - Gardasil 9 | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 High - HPV9 Low | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 Medium - HPV9 Low | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |
| HPV9 High - HPV9 Medium | XX | XX | (xx.x) | XX | XX | (xx.x) | XX.X | xx.x; | XX.X |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


N = Number of participants with available results who were seronegative (i.e, concentrations less than the LLOQ) at baseline

n (%) = number/percentage of participants with concentration equal or above specified value.

Seroconversion is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOQ) in the serum of participants seronegative before vaccination

#### Table 14.2.2.2

Differences of anti-HPV IgG Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - [Low, Med, High] and Gardasil9 group]

Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| <br>` ~ | ~ | <br><u>'</u> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | First | Study Group | Second | d Study Group | Di | fference |
| | | | N | n (%) | N | n (%) | % | 95% CI |

95% CI = 95% confidence interval computed based on Miettinen and Nurminen method. The concentration below the assay cut-off will be replaced by half the cut-off (LLOQ/2). Concentration above the ULOQ will be replaced by the ULOQ Programming Notes

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.2.2.3: Summary of anti-HPV Neutralizing Antibody GMTs and seropositivity for each antigen at Day 1, Month 2, Month 3 and Month 7 (Per Protocol Set)

GSK Vaccines

Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.2.2.3

Summary of anti-HPV Neutralizing Antibody GMTs and seropositivity for each antigen at Day 1, Month 2, Month 3 and Month 7

Per Protocol Set

| | Pre- | | | | | |
|---|---|---|---|---|---|---|
| | vaccination | | | | | |
| Visit | status | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 |
| Day 1 | Seronegative | N | xxx | XXX | xxx | XXX |
| | _ | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMT (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X.X | X.X | X.X | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMT | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | Seropositive | N | xxx | XXX | xxx | XXX |
| | _ | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMT (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X.X | x.x | x.x | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMT | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | N | xxx | xxx | xxx | xxx |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMT (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X.X | X.X | X.X | x.x |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMT | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


#### Table 14.2.2.3

Summary of anti-HPV Neutralizing Antibody GMTs and seropositivity for each antigen at Day 1, Month 2, Month 3 and
Month 7
Per Protocol Set

| Visit | Pre-<br>vaccination<br>status | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 |
|---|---|---|---|---|---|---|
| Month 2 | Seronegative | N | x | x | X | X |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | 95% CI seropositivity | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | GMT (GSD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | | Median | X . X | X • X | X.X | X.X |
| | | Min - Max | x - x | x - x | x - x | x - x |
| | | 95% CI GMT | x.x - x.x | x.x - x.x | x.x - x.x | x.x - x.x |
| | | n > ULOQ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | | | | | | |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMT = Geometric Mean Titer. GSD = Geometric Standard

Deviation. LLOQ = Lower Limit of Quantification. ULOQ = Upper Limit of Quantification.

 ${\tt N}$  = number of participants in the Per Protocol Set at each visit and pre-vaccination status.

n (%) = number/percentage of participants with titer equal or above LLOQ.

95% CI GMT = 95% confidence interval derived using the log10-transformed antibody titers.

Seronegative is defined as the situation where antibodies are not elevated (i.e, titers less than the LLOQ) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, titers greater than or equal to the LLOQ) in the serum of participants.

The titer below the LLOQ will be replaced by half the LLOQ (LLOQ/2). Titer above the ULOQ will be replaced by the ULOQ.

Programming Notes

Programming Notes

Output ID: IM0005

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.2.2.4.1: Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group) (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.4.1

Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group)

Per Protocol Set

| Antigen: xxx Pre- | (LLOQ = xx; ULOQ = xx; Unit = xx) | | | | | | |
|---|---|---|---|---|---|---|---|
| vaccination | | Н | IPV9 Group | Gard | dasil 9 Group | Group | GMT Ratio |
| status | | N | Adjusted GMT | N | Adjusted GMT | Value | 95% CI |
| Seronegative | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| beronegaerve | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | xx.x | xx | xx.x | xx.x | xx.x; xx.x |
| Seropositive | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | xx | XX.X | xx | XX.X | xx.x | xx.x; xx.x |
| Total | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | xx | XX.X | XX.X | xx.x; xx.x |
| Seronegative | anti-HPV Neutralizing titer at Month 7 | | | | | | |
| 3 | HPV9 High / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Low / Gardasil 9 | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


95% CI

#### Table 14.2.2.4.1

Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] divided by Gardasil 9 group) Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

Prevaccination HPV9 Group Gardasil 9 Group Group GMT Ratio Adjusted GMT status N Adjusted GMT Value

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMT = Geometric Mean Titer.

N = Number of participants with available results

The analysis is based on ANOVA model with log10 transformed anti-qE antibody titers values as response variable and the study group and country as fixed effects.

Seronegative is defined as the situation where antibodies are not elevated (i.e, titers less than the LLOO) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, titers greater than or equal to the LLOQ) in the serum of participants.

95% CI GMT = 95% confidence interval derived using the log-transformed antibody titers.

The titer below the LLOQ will be replaced by half the LLOQ (LLOQ/2). Titer above the ULOQ will be replaced by the

Programming Notes

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Output ID: IM0003

Author:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


## Table 14.2.2.4.2: Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between HPV Groups (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.4.2

Ratio of anti-HPV Neutralizing Antibody GMTs for each antigen at Month 3 and Month 7 between HPV Groups

Per Protocol Set

| Pre- | | | T' | | 1 0 | 9 | CME D |
|---|---|---|---|---|---|---|---|
| vaccination | | | First Group | | Second Group | | GMT Ratio |
| status | | N | Adjusted GMT | N | Adjusted GMT | Value | 95% CI |
| Seronegative | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | XX.X; XX.X |
| Seropositive | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| - | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | xx.x | xx.x; xx.x |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| Total | anti-HPV Neutralizing titer at Month 3 | | | | | | |
| | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| Seronegative | anti-HPV Neutralizing titer at Month 7 | | | | | | |
| - | HPV9 High / HPV9 Medium | XX | XX.X | XX | XX.X | xx.x | xx.x; xx.x |
| | HPV9 Medium / HPV9 Low | XX | XX.X | XX | XX.X | XX.X | xx.x; xx.x |
| | HPV9 High / HPV9 Low | XX | XX.X | XX | XX.X | xx.x | xx.x; xx.x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. GMT = Geometric Mean Titer.

N = Number of participants with available results

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


The analysis is based on ANOVA model with log10 transformed anti-gE antibody titers values as response variable and the study group and country as fixed effect.

Seronegative is defined as the situation where antibodies are not elevated (i.e, titers less than the LLOQ) in the serum of participants.

Seropositive is defined as the appearance of antibodies (i.e, titers greater than or equal to the LLOQ) in the serum of participants.

95% CI GMT = 95% confidence interval derived using the log-transformed antibody titers.

The titer below the LLOQ will be replaced by half the LLOQ (LLOQ/2). Titer above the ULOQ will be replaced by the ULOO.

Programming Notes

Programming Notes

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Output ID: IM0013


Table 14.2.2.5: Differences of anti-HPV Neutralizing Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group) (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.5

Differences of anti-HPV Neutralizing Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group) Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| | First | t Study Group | Secor | nd Study Group | Di | fference |
|---|---|---|---|---|---|---|
| | N | n (%) | N | n (%) | % | 95% CI |
| Seroconversion Rate at Month 3 | | | | | | |
| HPV9 High - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Medium - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Low - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 High - HPV9 Low | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Medium - HPV9 Low | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 High - HPV9 Medium | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| Seroconversion Rate at Month 7 | | | | | | |
| HPV9 High - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Medium - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Low - Gardasil 9 | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 High - HPV9 Low | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 Medium - HPV9 Low | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |
| HPV9 High - HPV9 Medium | XX | xx (xx.x) | XX | xx (xx.x) | XX.X | xx.x; xx |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author:

N = Number of participants with available results who were seronegative (i.e, concentrations less than the LLOQ) at

n (%) = number/percentage of participants with concentration equal or above specified value.

Seroconversion is defined as the appearance of antibodies (i.e, titers greater than or equal to the LLOQ) in the serum of participants seronegative before vaccination

#### Table 14.2.2.5

Differences of anti-HPV Neutralizing Antibody Seroconversion Rate for each antigen at Month 3 and Month 7 between Groups (HPV group [different potencies - Low, Med, High] and Gardasil9 group)

Per Protocol Set

Antigen: xxx (LLOQ = xx; ULOQ = xx; Unit = xx)

| · | Ι | First S | tudy Group | Second | l Study Group | Dif | ference |
|---|---|---------|------------|--------|---------------|-----|---------|
| | _ | N | n (%) | N | n (%) | % | 95% CI |

95% CI = 95% CI computed based on Miettinen and Nurminen method.

The titer below the LLOQ will be replaced by half the LLOQ (LLOQ/2). Titer above the ULOQ will be replaced by the ULOQ.

Programming Notes

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001) WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.2.2.6: Correlation between anti-HPV Immunoglobulin Antibody Concentration and anti-HPV Neutralizing Antibody Titers for each antigen at Day 1, Month 2, Month 3 and Month 7 (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.2.2.6

Correlation between anti-HPV Immunoglobulin Antibody Concentration and anti-HPV Neutralizing Antibody Titers for each antigen at Day 1, Month 2, Month 3 and Month 7

Per Protocol Set

Antigen: xxx

| | | | Pearson coefficie | ent of |
|-------------|---------|----|-------------------|---------|
| Study Dose | Visit | n | correlation | p-value |
| HDHO Hi wh | Da. 1 | | | • |
| HPV9 High | Day 1 | XX | X.XXX | 0.xxx |
| | Month 2 | XX | X.XXX | 0.xxx |
| | Month 3 | XX | X.XXX | 0.xxx |
| | Month 7 | XX | x.xxx | 0.xxx |
| | Overall | xx | x.xxx | 0.xxx |
| HPV9 Medium | Day 1 | xx | x.xxx | 0.xxx |
| | Month 2 | XX | x.xxx | 0.xxx |
| | Month 3 | XX | x.xxx | 0.xxx |
| | Month 7 | XX | x.xxx | 0.xxx |
| | Overall | XX | x.xxx | 0.xxx |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

n is the number of samples with both concentration and titer values.

Pearson correlation will be computed by the log10-transformation of the antibody concentration. Samples testing below the LLOQ or above the ULOQ in either assay were excluded from the analysis.

Programming Notes

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

Output ID: IM0007

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.2.2.7: Functional Relationship between the Assay Methods for each antigen (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| Study Dose | Visit | n | Intercept (95% CI for | |
|---|---|---|---|---|
| | | | Intercept) | Slope (95% CI for slope) |
| PV9-High | Day 1 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| , | Month 2 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Month 3 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Month 7 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Overall | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| PV9-Medium | Day 1 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Month 2 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Month 3 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Month 7 | xxx | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Overall | XXX | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| PV9-Low | | | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. ECL = Electrochemiluminescence assay. PBNA = Pseudovirion-Based Neutralization Assay

n is the number of samples with both concentration and titer values.

Deming's regression model is fitted to the Anti-HPV IgG antibody concentration (ECL) with Anti-HPV Neutralizing titers (PBNA) as a covariate.

Deming's regression will be computed by the log10-transformation of the antibody concentration and neutralizing titer. Samples testing below the LLOQ or above the ULOQ in either assay were excluded from the assay.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


### 

Antigen: xxx

| Study Dose | Visit | n | Intercept (95% CI for | |
|------------|-------|---|-----------------------|--------------------------|
| | | | Intercept) | Slope (95% CI for slope) |

Programming Notes

Output ID: IM0008

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\_213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.2.2.8 Summary of qualitative comparison between ECL and PBNA for each antigen by time point (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.2.2.8

Summary of qualitative comparison between ECL and PBNA for each antigen by time point Per Protocol Set

| | Antigen: | XXX | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study dose | Visit | n | Pos/<br>Pos | Neg/<br>Neg | Pos/<br>Neg | Neg/<br>Pos | IgG %<br>+ve | Neutralizing<br>titers % +ve | Agreement<br>rate % | Kappa | McNema<br>p-value | Kappa p-<br>value |
| study dose | VISIC | 11 | 103 | iveg | iveg | 105 | 100 | CICCIS 6 IVE | Tace o | карра | p value | varue |
| HPV9-High | Day 1 | XX | XX | XX | XX | XX | XX | XX | XX | xx | 0.xxx | 0.xxx |
| | Month 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Month 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Month 7 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Overall | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| HPV9-Medium | Day 1 | XX | XX | XX | XX | XX | XX | xx | XX | XX | 0.xxx | 0.xxx |
| | Month 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Month 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Month 7 | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |
| | Overall | XX | XX | XX | XX | XX | XX | XX | XX | XX | 0.xxx | 0.xxx |

HPV9-Low Gardasil 9 Total

Abbreviations: HPV = Human Papillomavirus. ECL = Electrochemiluminescence assay. PBNA = pseudovirion-based neutralization assay.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

n is the number of samples with both concentration and titer values are available.

Percentages are based on n.

Pos/Pos is the number of participants seropositive with both ECL and PBNA.

Neg/Neg is the number of participants seronegative with both ECL and PBNA.

Pos/Neg is the number of participants seropositive with ECL and seronegative with PBNA.

Neg/Pos is the number of participants seronegative with ECL and seropositive with PBNA.

Seronegative is defined as the situation where antibodies are not elevated (i.e, concentrations less than the LLOQ) in the serum of participants.

# $\hbox{ Table 14.2.2.8} \\ \hbox{Summary of qualitative comparison between ECL and PBNA for each antigen by time point } \\ \hbox{Per Protocol Set}$

Antigen: xxx

| | | | Pos/ | Neg/ | Pos/ | Neg/ | IgG % | Neutralizing | Agreement | | McNema | Kappa p- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study dose | Visit | n | Pos | Neg | Neg | Pos | +ve | titers % +ve | rate % | Kappa | p-value | value |

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to the LLOQ) in the serum of participants.

Programming Notes

Output ID: LS0014

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx




Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\
GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx




Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\
GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


05FEB2024 Version Date:
Table 14.3.1.1: Overall Summary of Grade 3 Solicited Administration Site Events and Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

Page X
GSK Vaccines

of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.1.1

Overall Summary of Grade 3 Solicited Administration Site Events and Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9<br>Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Any grade 3 solicited event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |
| Any grade 3 solicited administration site event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |
| Any grade 3 solicited systemic event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |

Source: Listing xx.x.x.x

Document:

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

 ${\tt N}$  is the number of participants in the Exposed Set for each period except Overall dose, where  ${\tt N}$  is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Data Lock Point.

MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

Output ID: SE0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Author:


Table 14.3.1.2.1: Number and Percentage of Participants of each Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Table 14.3.1.2.1

Number and Percentage of Participants of each Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one grade 3 | | | | | | |
| solicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| administration site event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Redness at injection site | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Swelling at injection site | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| At least one grade 3 solicited | | | | | | |
| administration site event leading to medical attention | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| Injection site pain | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Redness at injection site | n (%)<br>[95% CI] | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Swelling at injection site | n (%)<br>[95% CI] | [xx.x, xx.x]<br>x (x.x)<br>[xx.x, xx.x] | [xx.x, xx.x]<br>x (x.x)<br>[xx.x, xx.x] | [xx.x, xx.x]<br>x (x.x)<br>[xx.x, xx.x] | [xx.x, xx.x]<br>x (x.x)<br>[xx.x, xx.x] | [xx.x, xx.x]<br>x (x.x)<br>[xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


### Table 14.3.1.2.1

Number and Percentage of Participants of each Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | | | | |
|---------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

e is the number of events.

Author:

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


# Table 14.3.1.2.2: Summary of duration of Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.2.2

Summary of duration of Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall

Exposed Set

| Period: After first vaccine dose / After | second vaccine dose / | After third | vaccine dose | / Overall | (dose) | |
|---|---|---|---|---|---|---|
| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| Event | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| T. 1 | | | | | | |
| Injection Site Pain | n | X | X | X | X | X |
| | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | X.X | X • X | X . X | X . X | X . X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Redness at Injection Site | n | х | х | Х | x | Х |
| • | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | X.X | X . X | x.x | X.X | X.X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Swelling at Injection Site | n | Х | Х | х | Х | X |
| ewelling do injection site | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | x.x | X.X | x.x | X.X | X.X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.3.1.2.2

Summary of duration of Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

| Period: After first vaccine dose / Af | ter second vaccine dose / | After third | vaccine dose | / Overall | (dose) | |
|---|---|---|---|---|---|---|
| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| Event | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

Programming Notes

Output ID: DUR0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Version Date:

05FFB2024

Table 14.3.1.2.3: Number and percentage of participants with Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

## Table 14.3.1.2.3

Number and percentage of participants with Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration Exposed Set

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Injection Site Pain | | | | | | |
| N* | | x | Х | Х | X | Х |
| 1 day | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 2 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 3 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 4 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=5 days | n (응) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Redness at Injection Site | | | | | | |
| N* | | x | Х | Х | X | Х |
| 1 day | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 2 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 3 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 4 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=5 days | n (응) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Swelling at Injection Site | e | | | | | |
| N* | | X | X | X | Х | х |
| 1 day | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 2 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 3 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 4 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=5 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Table 14.3.1.2.3

Number and percentage of participants with Grade 3 Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration

Exposed Set

| Period: After first vaccine do | se / After second s | vaccine dose / Af | ter third vaccine | dose / Overall | (participant) |
|---|---|---|---|---|---|
| | HPV9 | High HPV9 Me | dium HPV9 Low | Gardasil 9 | 9 Total |
| | (N=XX | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

Source: Listing xx.x.x.x

Author:

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

 $N^*$  is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs

n is the number of participants with a specified duration of an event

Percentages are calculated as 100 \* n/N\*.


Table 14.3.1.3.1: Number and Percentage of Participants of each Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Table 14.3.1.3.1

Number and Percentage of Participants of each Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| At least one grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| solicited systemic event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Fever | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Headache | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Myalgia | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Arthralgia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Fatigue | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| At least one grade 3 | | | | | | |
| solicited systemic event | (0) | | | , , | | , , |
| leading to medical attention | n (%) | | x (x.x) | | x (x.x) | x (x.x) |
| | [95% CI] e<br>n (%) | [XX.X, XX.X] X<br>X (X.X) | [xx.x, xx.x] x<br>x (x.x) | [XX.X, XX.X] X<br>X (X.X) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) |
| Fever | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Headache | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Mara I ari a | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Myalgia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Arthralgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Table 14.3.1.3.1

Number and Percentage of Participants of each Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Fatigue | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

e is the number of events.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson


# Table 14.3.1.3.2: Summary of duration of Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.3.2

Summary of duration of Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| Event | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Fever | | | | | | |
| Level | n<br>Mean (SD) | x<br>x.x (x.xx) | x<br>x.x (x.xx) | x<br>x.x (x.xx) | x<br>x.x (x.xx) | x<br>x.x (x.xx) |
| | Median | X . X | X.X | X • X | X.X | X • X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Headache | n | x | х | х | x | Х |
| | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | X.X | X.X | X.X | X.X | X.X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Myalgia | n | x | Х | Х | Х | х |
| 11101910 | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | X.X | X.X | x.x | x.x | x.x |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| not be a lesi a | | | | | | |
| Arthralgia | n | X | X | X | X | X |
| | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| | Median | X.X | X.X | X.X | X.X | X.X |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | X - X |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |
| Fatigue | n | Х | x | х | x | Х |
| | Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

## Table 14.3.1.3.2

Summary of duration of Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| Event | Statistic | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| | Median | x.x | х.х | x.x | x.x | х.х |
| | Q1 - Q3 | x - x | x - x | x - x | x - x | x - x |
| | Min - Max | x - x | x - x | x - x | x - x | x - x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Programming Notes

Output ID: DUR0001

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.3.1.3.3: Number and percentage of participants with Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration (Exposed Set)

GSK Vaccines

Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.3.3

Number and percentage of participants with Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (participant) HPV9 High HPV9 Medium HPV9 Low Gardasil 9 Total (N=XXX)(N=XXX)(N=XXX)(N=XXX)(N=XXX)Fever Ν\* Х Х Х Х Х 1 day n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)2 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)3 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)4 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)>=5 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)Headache Ν\* Х Х Х Х Х 1 day n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)2 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)3 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)4 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)>=5 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)Myalqia Ν\* Х х х х х 1 day n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)2 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)3 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)4 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)>=5 days n (%) x (x.x)x (x.x)x (x.x)x (x.x)x (x.x)

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

Table 14.3.1.3.3

Number and percentage of participants with Grade 3 Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by days of duration

Exposed Set

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Arthalgia | | | | | | |
| N* | | Х | X | Х | X | Х |
| 1 day | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 2 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 3 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 4 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=5 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Fatigue | | | | | | |
| N* | | X | X | X | X | X |
| 1 day | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 2 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 3 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 4 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| >=5 days | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

 $N^*$  is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs

n is the number of participants with a specified duration of an event

Percentages are calculated as 100 \*  $n/N^*$ .


Author:


# Table 14.3.1.4: Summary of Participants with any Grade 3 Unsolicited Events and Serious Adverse Events (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one Grade 3<br>Unsolicited Adverse Event | n (%)<br>[95% CI] e | | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one causally<br>related Grade 3 Unsolicited<br>Adverse Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one Serious Adverse<br>Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one causally<br>related Serious Adverse<br>Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one fatal Serious<br>Adverse Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one causally<br>related fatal Serious<br>Adverse Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

# 

| Period: After first vaccine | lose / After second vaccin | e dose / After | third vaccine dos | se / Overall (d | ose) / Overall | (participant) |
|---|---|---|---|---|---|---|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total | |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

e is the number of events.

Includes AEs with an onset date on or after the date of first vaccine up to Study End.

95% CI are based on Clopper-Pearson

Causally related events are those that are related to HPV vaccine according to the investigator.

The unsolicited adverse event summaries include events that are reported within 28 days (Day 1 - 28) after each

vaccine dose. The serious adverse event summaries include events that are reported upto Study End.

MedDRA version xx.x.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx

Author:


Table 14.3.1.5: Number and Percentage of Participants of each Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.1.5

Number and Percentage of Participants of each Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| · | · | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| At least one grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| unsolicited adverse event | [95% CI] e | | [xx.x, xx.x] x | | | |
| < <system 1="" class="" organ="">&gt;</system> | n (%) | | | x (x.x) | | x (x.x) |
| < <pre>&lt;<pre>ferred term 1&gt;&gt;</pre></pre> | [95% CI] e<br>n (%) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) |
| //rreferred term 1// | [95% CI] e | [xx.x, xx.x] x | | [xx.x, xx.x] x | | [xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | , , |
| //Custom summa slage 222 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 2="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 1&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| ( TICICIICA CCIM 1// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 2&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Colored Celm 2// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx

Author:


3.0

### Table 14.3.1.5

Number and Percentage of Participants of each Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | | | | |
|---------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

Author:

95% CI are based on Clopper-Pearson

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


3.0

Table 14.3.1.6: Number and Percentage of Participants of causally related Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Vaccine: HPV

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.1.6

Number and Percentage of Participants of causally related Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| <b>Уриготограно</b> | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one causally related | | | | | | |
| grade 3 unsolicited adverse | n (2) | v (v v) | x (x.x) | v (v v) | v (v v) | x (x.x) |
| event | [95% CI] e | | [xx.x, xx.x] x | | | |
| | [300 01] 6 | [MAIN, MAIN] A | [M.M, M.M] M | [111.11] 11.11] 11 | [M.M, M.M] A | [22.27] 22.21] 22 |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system (="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <pre></pre> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x]x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 2&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| (\Frederical telm 2// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| //Custom support slags 222 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 2="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 1&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| //irerefred cerm 1// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 2="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| VIICICIICA CEIM 2// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Table 14.3.1.6

Number and Percentage of Participants of causally related Grade 3 Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|-----------|-------------|----------|------------|---------|
| (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYY

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


# Table 14.3.1.7: Number and Percentage of Participants of Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.7

Number and Percentage of Participants of Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one serious | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| adverse event | | [xx.x, xx.x] x | | [xx.x, xx.x] x | , , | , , |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | , , | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>erred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | , , | , , | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | , , |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term. e is the number of events; participants with events in more than one preferred term are counted once in each of

those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Data Lock Point.

95% CI are based on Clopper-Pearson

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.3.1.7

Number and Percentage of Participants of Serious Adverse Events Reported up to Study End by System Organ Class and
Preferred Term
Exposed Set

| HPV9 | птин п | irvə Mediulli - r | HPV9 Low | Gardasil 9 | Total |
|------|--------|-------------------|----------|------------|---------|
| | XX) ( | N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\_213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


# Table 14.3.1.8: Number and Percentage of Participants of causally related Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.8

Number and Percentage of Participants of causally related Serious Adverse Events Reported up to Study End by System
Organ Class and Preferred Term
Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one causally related serious adverse event | | | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | | , , |
| < <pre>&lt;<pre>erred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | , , |
| < <system 1="" class="" organ="">&gt; &lt;<preferred 1="" term="">&gt;</preferred></system> | n (%)<br>[95% CI] e<br>n (%)<br>[95% CI] e | x (x.x) [xx.x, xx.x] x x (x.x) [xx.x, xx.x] x | [xx.x, xx.x] x<br>x (x.x) | x (x.x) [xx.x, xx.x] x x (x.x) [xx.x, xx.x] x | [xx.x, xx.x] x<br>x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Study End.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.3.1.8

Number and Percentage of Participants of causally related Serious Adverse Events Reported up to Study End by System
Organ Class and Preferred Term
Exposed Set

| HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|-----------|-------------|----------|------------|---------|
| (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

95% CI are based on Clopper-Pearson Causally related events are those that are related to HPV vaccine according to the investigator. MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749\) (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\\\ 213749\(\text{HPV9-AS04-001}\) \(\text{WZA97329}\) TFL\Shells\\\\ \V3.0\\\_05FEB2024.docx\)


# Table 14.3.1.9: Number and Percentage of Participants of fatal Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.9

Number and Percentage of Participants of fatal Serious Adverse Events Reported up to Study End by System Organ

Class and Preferred Term

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one fatal serious | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| adverse event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| //Creaton oncen along 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 1="" class="" organ="">&gt; "[9</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| ((ITELETIEG CEIM 1)) | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 2="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Vileteffed telm 2// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <system 1="" class="" organ="">&gt;</system> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Coystem Organ Class 1// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| //Lielelied felw 1// | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Study End.

95% CI are based on Clopper-Pearson

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


## Table 14.3.1.9

Number and Percentage of Participants of fatal Serious Adverse Events Reported up to Study End by System Organ
Class and Preferred Term
Exposed Set

| НР | va urdu t | HPV9 Mealum 1 | HPV9 Low | Gardasil 9 | Total |
|-----|-----------|---------------|----------|------------|---------|
| (N= | =XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\_213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.3.1.10: Number and Percentage of Participants of causally related fatal Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.1.10

Number and Percentage of Participants of causally related fatal Serious Adverse Events Reported up to Study End by System Organ Class and Preferred Term

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one causally | | | | | | |
| related fatal serious | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| adverse event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| //Cusham suman slass 1>> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 1="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 1&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <pre></pre> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| ((D)) = 6 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <preferred 2="" term="">&gt;</preferred> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| //Custom support slags 122 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 1="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| //Lielelied felm 1>> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term. e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


## Table 14.3.1.10

Number and Percentage of Participants of causally related fatal Serious Adverse Events Reported up to Study End by

System Organ Class and Preferred Term

Exposed Set

| 1 | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|-----------|-------------|----------|------------|---------|
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

Includes AEs with an onset date on or after the date of first vaccine up to Study End. 95% CI are based on Clopper-Pearson

Causally related events are those that are related to HPV vaccine according to the investigator. MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Author:


# Table 14.3.1.11: Number and Percentage of Participants of Laboratory Parameters Outside normal range at Day 7 after the first vaccine dose (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Biochemical | | | | | | |
| < <lab 1="" parameter="">&gt;</lab> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| < <lab 2="" parameter="">&gt;</lab> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| < <lab 3="" parameter="">&gt;</lab> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Hematological | | | | | | |
| < <lab 1="" parameter="">&gt;</lab> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


Author:


Table 14.3.2.1: Overall Summary of Solicited Administration Site Events and Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

Page X
GSK Vaccines

of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.2.1

Overall Summary of Solicited Administration Site Events and Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9<br>Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total (N=XXX) |
|---|---|---|---|---|---|---|
| Any solicited event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |
| Any solicited administration site event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |
| Any solicited systemic event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, | [xx.x, | [xx.x, | [xx.x, xx.x] | [xx.x, xx.x] |
| | e | xx.x] x | xx.x] x | xx.x] x | x | x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

 ${\tt N}$  is the number of participants in the Exposed Set for each period except Overall dose, where  ${\tt N}$  is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson


# GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Data Lock Point.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

Table 14.3.2.2: Number and Percentage of Participants of Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Table 14.3.2.2

Number and Percentage of Participants of each Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High (N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one solicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| administration site event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Redness at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Swelling at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| At least one solicited administration site event | n (%) | ( | () | () | ( | () |
| leading to medical attention | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Redness at injection site | n (%)<br>[95% CI] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Swelling at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

### Table 14.3.2.2

Number and Percentage of Participants of each Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| _ (parerelpane) | | | | | |
|---|---|---|---|---|---|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

e is the number of events.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


# Table 14.3.2.3: Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

## Table 14.3.2.3

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| At least one solicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| administration site event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Fever | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Headache | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| | u (%) | [xx.x, xx.x]<br>x (x.x) | [ xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) |
| Myalgia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| 7 11 7 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Arthralgia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Fatigue | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| racigue | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| At least one solicited | | | | | | |
| administration site event | | | | | | |
| leading to medical attention | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| reading to medical accention | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Fever | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Headache | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) | [xx.x, xx.x]<br>x (x.x) |
| Myalgia | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Arthralgia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Table 14.3.2.3

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Fatigue | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

e is the number of events.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson


Table 14.3.2.4: Number and Percentage of Participants of Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Table 14.3.2.4

Number and Percentage of Participants of each Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one solicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| administration site event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Redness at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Swelling at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author: Version Date: 05FFB2024
Table 14.3.2.4

Number and Percentage of Participants of each Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| At least one solicited administration site event | n (%) | ( | () | () | () | () |
| leading to medical attention | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Redness at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Swelling at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0


#### Table 14.3.2.4

Number and Percentage of Participants of each Solicited Administration Site Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (1 1 ) | | | | | |
|--------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

e is the number of events.

Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


Table 14.3.2.5: Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.5

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| At least one solicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| systemic event | [95% CI] e | | [xx.x, xx.x] x | | | |
| Fever | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 1 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 2 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 3 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Headache | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 1 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 2 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 3 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Myalgia | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 1 | n (%)<br>[95% CI] | x (x.x)<br>[xx.x, xx.x] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.3.2.5

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Arthralgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Fatigue | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| At least one solicited | | | | | | |
| systemic event leading to medical attention | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Fever | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Headache | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.3.2.5

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| | ~ (%) | () | () | () | () | () |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 3 | n (%)<br>[95% CI] | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Myalgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 5_5.5.5 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Arthralgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| iii ciii aigia | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Glade 1 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| Date faces | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Fatigue | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| C1 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 1 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| G | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |
| | n (응) | x (x.x) | | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

#### Table 14.3.2.5

Number and Percentage of Participants of Solicited Systemic Events Reported within 7 days (Days 1-7) after each vaccine dose and overall by Severity

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | | | | |
|---------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

e is the number of events. Percentages are calculated as 100 \* n/N.

95% CI are based on Clopper-Pearson

Output ID: SE0002

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\\GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


# Table 14.3.2.6.1: Solicited Events, Completeness Analysis, by Administration Site and Systemic Category by Intervention Group and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.6.1
Solicited Events, Completeness Analysis, by Administration Site and Systemic Category by Intervention Group and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Any solicited administration | . (0) | ( | ( | ( | () | ( |
| site event | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Injection site pain | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Redness at injection site | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Swelling at injection site | n (%)<br>[95% CI] | x (x.x) | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] | x (x.x)<br>[xx.x, xx.x] |
| Any solicited systemic event | n (%) | | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Fever | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Headache | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Myalgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Arthralgia | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |
| Fatigue | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] | [xx.x, xx.x] |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


#### Table 14.3.2.6.1

Solicited Events, Completeness Analysis, by Administration Site and Systemic Category by Intervention Group and overall

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|-----------|-------------|----------|------------|---------|
| (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

Source: Listing xx.x.x.x

Document:

Author:

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with documented absence or presence of the event on at least one day. Percentages are calculated as 100  $^{\star}$  n/N.

95% CI are based on Clopper-Pearson

[Source:  $\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM$ 


# Table 14.3.2.6.2: eDiary Collection, Compliance and Completeness in Solicited Events by Intervention Group and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.6.2 eDiary Collection, Compliance and Completeness in Solicited Events by Intervention Group and overall Exposed Set

| | | HPV9 High | | HP' | V9 Medium | F | HPV9 Low | Ga | ırdasil 9 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | | N | | N | | N | | N | |
| Solicited administration site | | | | | | | | | | | |
| event | | | | | | | | | | | |
| Injection site pain | | | | | | | | | | | |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX | x x (x.x |
| Doduces of inication site | 27.1 | | , | | , | | , | | | | , |
| Redness at injection site | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.) |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.) |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.: |
| Swelling at injection site | N* n (%) | xxx | x x (x.x) | xxx | x x (x.x) | xxx | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |
| Day 4 | N* n (%) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | xxx | x x (x.x) | XXX | $x \times (x.x)$ | XXX | x x (x.2 |
| Solicited systemic event | | | | | | | | | | | |
| Fever | | | | | | | | | | | |
| Day 1 | N* n (%) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX | x x (x.: |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x. |

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Table 14.3.2.6.2
eDiary Collection, Compliance and Completeness in Solicited Events by Intervention Group and overall
Exposed Set

| | | Н | PV9 High | HP' | V9 Medium | F | HPV9 Low | Gardasil 9 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | N | | N | | N | | N | N | |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x. |
| Day 4 | N* n (%) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x. |
| Headache | N* n (%) | xxx | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x. |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX X X (X. | x) xxx | x x (x. |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX X X (X. | XXX XXX | x x (x. |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX X X (X. | x) xxx | x x (x. |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x |
| Myalgia | N* n (%) | xxx | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x |
| Day 1 | N* n (%) | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX | $x \times (x.x)$ | XXX x x (x. | x) xxx | x x (x |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX X X (X. | x) xxx | x x (x |
| Day 3 | N* n (응) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | x) xxx | x x (x |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x |
| Arthralgia | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | xxx x x (x. | x) xxx | x x (x |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX X X (X. | xxx xxx | x x (x |
| Day 2 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | x) xxx | х х (х |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | $x \times (x.x)$ | XXX X X (X. | xxx xxx | x x (x |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | x) xxx | х х (х |
| Fatique | N* n (%) | xxx | x x (x.x) | xxx | x x (x.x) | xxx | x x (x.x) | XXX X X (X. | x) XXX | х х (х |
| Day 1 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | / | x x (x |
| Day 2 | N* n (%) | xxx | x x (x.x) | xxx | x x (x.x) | xxx | x x (x.x) | XXX X X (X. | / | x x (x |
| Day 3 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | / | x x (x |
| Day 4 | N* n (%) | XXX | x x (x.x) | XXX | x x (x.x) | XXX | x x (x.x) | XXX X X (X. | / | x x (x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

#### Table 14.3.2.6.2

eDiary Collection, Compliance and Completeness in Solicited Events by Intervention Group and overall Exposed Set

| Period: After first vaccine dose | After second vaccine | dose / After third | vaccine dose / Overa | ll (dose) / Overall | (participant) |
|---|---|---|---|---|---|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | N | N | N | N | N |

 $N^*$  is the number of participants with documented absence or presence of the event on that day. n is the number of participants with documented presence of the event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where there is documented presence of the event. Percentages are calculated as  $100 * n/N^*$ 

Programming Notes
All events will go up to day 7.

Output ID: SE0005

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.3.2.7.1: Summary of Participants with any Unsolicited Adverse Events and Potential Immune-Mediated Disease (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.7.1

Summary of Participants with any Unsolicited Adverse Events and Potential Immune-Mediated Disease Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one Unsolicited<br>Adverse Event | | | x (x.x)<br>[xx.x, xx.x] x | | | |
| At least one causally related Unsolicited Adverse Event | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one Unsolicited<br>Adverse Event Leading to<br>Medical Attention | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one Potential<br>Immune-Mediated Disease | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |
| At least one causally<br>related Potential Immune-<br>Mediated Disease | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | | |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval.

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

e is the number of events.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


#### Table 14.3.2.7.1

Summary of Participants with any Unsolicited Adverse Events and Potential Immune-Mediated Disease Exposed Set

| Period: | After f | first | vaccine | dose / | After | second | vaccine | dose / | After | third | vaccine | dose | / Overall | (dose) | / Overall | (participant) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | HPV9 | High | HPV9 | Mediu | m i | HPV9 Low | | Gardasil | 9 | Total | |
| | | | | | | (N=X) | XX) | (N=X) | XX) | | (N=XXX) | | (N=XXX) | | (N=XXX) | |

The unsolicited adverse event summaries include events that are reported within 28 days (Day 1 - 28) after each vaccine dose. The Potential Immune-Mediated Disease summaries include events that are reported upto Study End.

95% CI are based on Clopper-Pearson Causally related events are those that are related to HPV vaccine according to the investigator. MedDRA version xx.x.

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Document:

Version Number: 3.0 Author: Version Date: 05FFB2024

Table 14.3.2.7.2: Number and Percentage of Participants of Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.2.7.2

Number and Percentage of Participants of Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one unsolicited adverse event | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | , , | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <system 2="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | , , | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>erred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | x (x.x) | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx

Author:


3.0

#### Table 14.3.2.7.2

Number and Percentage of Participants of Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | | | | |
|---------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

Document:

Author:

95% CI are based on Clopper-Pearson

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


Table 14.3.2.7.3: Number and Percentage of Participants of causally related Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.2.7.3

Number and Percentage of Participants of causally related Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one causally related unsolicited adverse event | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x | |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x]x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>c<preferred 2="" term="">&gt;</preferred></pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <system 2="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 1&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <pre>&lt;<pre>erred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | | x (x.x) | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


#### Table 14.3.2.7.3

Number and Percentage of Participants of causally related Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (parerelpane) | | | | | |
|---------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYY

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


Table 14.3.2.7.4: Number and Percentage of Participants with Unsolicited Adverse Events Leading to Medical Attention Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.2.7.4

Number and Percentage of Participants with Unsolicited Adverse Events Leading to Medical Attention Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one unsolicited | n (%) | v (v v) | x (x.x) | v (v v) | v (v v) | v (v v) |
| adverse event | [95% CI] e | , , | [xx.x, xx.x] x | | | |
| < <system 1="" class="" organ="">&gt;</system> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <pre></pre> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 1&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <pre></pre> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x]x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>ferred term 2&gt;&gt;</pre></pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre></pre></pre></pre></pre></pre></pre> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| //Cusham suman slass 2>> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 2="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| ((D) - 6 1 + 1 > . | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <preferred 1="" term="">&gt;</preferred> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 2="" term="">&gt;</preferred> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx

Author:


3.0

#### Table 14.3.2.7.4

Number and Percentage of Participants with Unsolicited Adverse Events Leading to Medical Attention Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class and Preferred Term Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| (Parerpane) | | | | | |
|-------------|-----------|-------------|----------|------------|---------|
| | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

95% CI are based on Clopper-Pearson

 $[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] \ IQVIA \ DDMMMYY \quintiles.$ 

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


Version Date:

05FFB2024

Table 14.3.2.7.5: Number and Percentage of Participants with Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class, Preferred Term and Severity (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Table 14.3.2.7.5

Number and Percentage of Participants with Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class, Preferred Term and Severity Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| At least one unsolicited | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| adverse event | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Glade 1 | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | [95% CI] e | | [xx.x, xx.x] x | | [xx.x, xx.x] x | |
| Grade 3 | n (%) | x (x.x) | | x (x.x) | x (x.x) | x (x.x) |
| 01440 0 | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 1="" class="" organ="">&gt;</system> | [95% CI] e | | [xx.x, xx.x] x | | | |
| Consider 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade I | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Crado 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Glade 5 | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>ferred term 1&gt;&gt;</pre> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| VIICICIICA CCIM 177 | [95% CI] e | [xx.x, xx.x] x | | | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 01440 1 | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Grade 2 | n (응) | x (x.x) | | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | | [xx.x, xx.x] x | | | |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document:

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


3.0

Table 14.3.2.7.5

Number and Percentage of Participants with Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class, Preferred Term and Severity

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall

(participant)

| | | HPV9 High (N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| - | | (IN-VVV) | (N-XXX) | (IV-XXX) | (N-VVV) | (N-VVV) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <pre>&lt;<pre>referred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Mild | [95% CI] e | [xx.x, xx.x] x | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Moderate | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| _ | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Severe | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | | |
| ((Custom summer slage 2)) | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| < <system 2="" class="" organ="">&gt;</system> | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Mild | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| MIIQ | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Moderate | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Moderate | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Severe | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Severe | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| (VIICICIICA CCIM 1// | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Mild | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 11114 | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Moderate | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| 110 401 400 | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Severe | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| < <preferred 2="" term="">&gt;</preferred> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Mild | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [xx.x, xx.x] x | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x |
| Moderate | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | |
| Severe | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | [95% CI] e | [XX.X, XX.X] X | [xx.x, xx.x] x | [xx.x, xx.x] x | [xx.x, xx.x] x | [XX.X, XX.X] X |

Source: Listing xx.x.x.x

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author: Version Number:

#### Table 14.3.2.7.5

Number and Percentage of Participants with Unsolicited Adverse Events Reported within 28 days (Days 1-28) after each vaccine dose and overall by System Organ Class, Preferred Term and Severity

Exposed Set

Period: After first vaccine dose / After second vaccine dose / After third vaccine dose / Overall (dose) / Overall (participant)

| HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
|-----------|-------------|----------|------------|---------|
| (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set for each period except Overall dose, where N is the total number of doses in the Exposed Set.

n is the number of participants with an event in the Exposed Set for each period except Overall dose, where n is the total number of doses in the Exposed Set where an event occurs.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Unsolicited AEs include serious AEs.

MedDRA version xx.x.

95% CI are based on Clopper-Pearson

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYY

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


## Table 14.3.2.8.1: Number and Percentage of Participants of Potential Immune-Mediated Disease Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.8.1

Number and Percentage of Participants of Potential Immune-Mediated Disease Reported up to Study End by System Organ

Class and Preferred Term

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one potential | n (%) | v (v v) | x (x.x) | v (v v) | x (x.x) | v (v v) |
| immune-mediated disease | | [xx.x, xx.x] x | | [xx.x, xx.x] x | | |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | , , | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | |
| < <pre>&lt;<pre>erred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x) | | x (x.x) |
| < <system 1="" class="" organ="">&gt;</system> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | , , | | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x |
| < <preferred 1="" term="">&gt;</preferred> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x)<br>[xx.x, xx.x] x | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term. e is the number of events; participants with events in more than one preferred term are counted once in each of

those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Study End.

95% CI are based on Clopper-Pearson

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


#### Table 14.3.2.8.1

Number and Percentage of Participants of Potential Immune-Mediated Disease Reported up to Study End by System Organ

Class and Preferred Term

Exposed Set

| HPV9 H | igh HPV9 Med: | | Gardasil 9 | Total |
|--------|---------------|---------|------------|---------|
| (N=XXX | | (N=XXX) | (N=XXX) | (N=XXX) |

MedDRA version xx.x.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


Table 14.3.2.8.2: Number and Percentage of Participants with causally related Potential Immune-Mediated Disease Reported up to Study End by System Organ Class and Preferred Term (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.8.2

Number and Percentage of Participants with causally related Potential Immune-Mediated Disease Reported up to Study

End by System Organ Class and Preferred Term

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one potential | n (%) | x (x x) | x (x.x) | y (y y) | x (x.x) | x (x x) |
| immune-mediated disease | ٠, | [xx.x, xx.x] x | , , | [xx.x, xx.x] x | , , | ' ' |
| < <system 1="" class="" organ="">&gt;</system> | n (%) | | , , | | x (x.x) | |
| | [95% CI] e<br>n (%) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | [xx.x, xx.x] x<br>x (x.x) | |
| < <preferred 1="" term="">&gt;</preferred> | [95% CI] e | [xx.x, xx.x] x | . , . | | [xx.x, xx.x] x | |
| < <pre>&lt;<pre>referred term 2&gt;&gt;</pre></pre> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | | x (x.x)<br>[xx.x, xx.x] x |
| < <system 1="" class="" organ="">&gt;</system> | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| (15) Stem Olgan Class 1// | [95% CI] e | [xx.x, xx.x] x | | | [xx.x, xx.x] x | |
| < <preferred 1="" term="">&gt;</preferred> | n (%)<br>[95% CI] e | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | x (x.x)<br>[xx.x, xx.x] x | | ' ' |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus. CI = Confidence Interval. MedDRA = Medical dictionary for regulatory activities

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

Participants with multiple events in the same preferred term are counted only once in that preferred term.

e is the number of events; participants with events in more than one preferred term are counted once in each of those preferred terms.

Includes AEs with an onset date on or after the date of first vaccine up to Study End.

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


#### Table 14.3.2.8.2

Number and Percentage of Participants with causally related Potential Immune-Mediated Disease Reported up to Study

End by System Organ Class and Preferred Term

Exposed Set

| HPV9 H | igh HPV9 Med: | | Gardasil 9 | Total |
|--------|---------------|---------|------------|---------|
| (N=XXX | | (N=XXX) | (N=XXX) | (N=XXX) |

95% CI are based on Clopper-Pearson MedDRA version xx.x.

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


### Table 14.3.2.9.1: Number and Percentage of Participants of Pregnancies Reported up to Study End (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.2.9.1 Number and Percentage of Participants of Pregnancies Reported up to Study End Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low<br>(N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one pregnancy reported during the study | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

N is the number of participants in the Exposed Set.

n is the number of participants included in each category.

Percentages are calculated as 100 \* n/N.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


# Table 14.3.2.9.2: Number and Percentage of Participants of Pregnancies Reported around each Vaccination (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| | | HPV9 High<br>(N=XXX) | HPV9 Medium (N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total (N=XXX) |
|---|---|---|---|---|---|---|
| At least one pregnancy reported around first vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least one pregnancy reported around second vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least one pregnancy reported around third vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Percentages are calculated as 100 \* n/N.

Around each vaccination is defined as any pregnancy reported within 30 days before and 45 days after each vaccination.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


# Table 14.3.2.9.3: Number and Percentage of Participants of Pregnancies Outcomes Reported up to Study End (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of pregnancies reported | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least one pregnancy reported around first | | | | | | |
| vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Outcome: | | | | | | |
| Live infant, no apparent congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Live infant congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Elective termination, no apparent congenital | | | | | | |
| anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Elective termination congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Spontaneous abortion, no apparent congenital | | | | | | |
| anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Spontaneous abortion congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Stillbirth, no apparent congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Stillbirth congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Ectopic pregnancy | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Molar pregnancy | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Lost to follow-up | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Pregnancy ongoing | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least one pregnancy reported around second | | | | | | |
| vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Live infant, no apparent congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Document:

\\quintiles.net\Enterprise\Apps\sasdata\SAS\\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


3.0

Table 14.3.2.9.3

Number and Percentage of Participants of Pregnancies Outcomes Reported up to Study End

Exposed Set

| | | HPV9 High<br>(N=XXX) | HPV9 Medium<br>(N=XXX) | HPV9 Low (N=XXX) | Gardasil 9<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| At least one pregnancy reported around third | | | | | | |
| vaccination | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Live infant, no apparent congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| At least one pregnancy reported around all | | | | | | |
| vaccinations | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Live infant, no apparent congenital anomaly | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Percentages are calculated as 100 \* n/N.

Around each vaccination is defined as any pregnancy reported within 30 days before and 45 days after each vaccination.

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


### Table 14.3.3.1: Summary of Laboratory Parameters Grades: Hematology by study group and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Table 14.3.3.1

Summary of Laboratory Parameters Grades: Hematology by study group and overall Exposed Set

| Lab parameter | | | | | | |
|---|---|---|---|---|---|---|
| Visit | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| Grade | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Hemoglobin | | | | | | |
| Visit 1 | | | | | | |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 4 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 2 | | | | | | |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 4 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Percentages are calculated as 100 \* n/N.

Baseline is the result at Visit 1.

See table 13 in the protocol for definition of the grades for each lab parameter

Programming note:

Include hemoglobin, hemoglobin change from baseline, white blood cells increase, white blood cell decrease, lymphocyte decrease, neutrophils decrease, eosinophils and platelet decrease

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Table 14.3.3.2: Summary of Laboratory Parameters Grades: Chemistry by study group and overall (Exposed Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

| Lab parameter | | | | | | |
|---|---|---|---|---|---|---|
| Visit | | HPV9 High | HPV9 Medium | HPV9 Low | Gardasil 9 | Total |
| Grade | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Blood Urea Nitrogen | | | | | | |
| Visit 1 | | | | | | |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 4 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Visit 2 | | | | | | |
| Grade 1 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 2 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 3 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Grade 4 | n (%) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source: Listing xx.x.x.x

Abbreviations: HPV = Human Papillomavirus.

Percentages are calculated as 100 \*n/N.

See table 13 in the protocol for definition of the grades for each lab parameter

Programming note:

Include blood urea nitrogen, AST and ALT

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Filename.sas] IOVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


Figure 16.1.2.1: Reverse Cumulative Curve (RCC) for anti-HPV IgG Antibody Concentration for each antigen at Day 1, Month 2, Month 3, Month 7 and Month 12 (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Figure 16.1.2.1

Reverse Cumulative Curve (RCC) for anti-HPV IgG Antibody Concentration for each antigen at Day

1, Month 2, Month 3, Month 7 and Month 12

Per Protocol Set

Antigen: xx (LLOQ=xx; ULOQ=xx; Unit=xx) Timepoint: Day 1/Month 2/Month 3/Month 7/Month 12



 $\begin{array}{l} \textit{Programming Notes} \\ \textbf{The above graph is for reference and following programming notes should be followed} \\ \end{array}$ 

Document:

Author:


Version Date:

05FEB2024

### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

- 1. Represent number of participants in percentage on y-axis and log of the concentration value on x-axis
- 2. Present separate curve for each treatment group. Present separate plots for each timepoint and antigen

Output ID: IM0011

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


Author:


Figure 16.1.2.2: Reverse Cumulative Curve (RCC) for anti-HPV Neutralizing Antibody Titers for each antigen at Day 1, Month 2, Month 3 and Month 7 (Per Protocol Set)

Figure 16.1.2.2

Reverse Cumulative Curve (RCC) for anti-HPV Neutralizing Antibody Titers at Day 1, Month 2, Month 3 and Month 7

Exposed Set

IM0012: This output uses shell IM0011 [Figure 16.1.2.1]

#### Programming Notes

• Replace footnotes in original shell with those listed above

Figure 16.1.2.3: Scatterplot for Deming's regression of the Anti-HPV Neutralizing titers and Anti-HPV IgG antibody concentrations for each antigen (Per Protocol Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Figure 16.1.2.3

Scatterplot for Deming's regression of the Anti-HPV Neutralizing titers and Anti-HPV IgG antibody concentrations for each antigen

Per Protocol Set



Source: Listing xx.x.x.x

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749\) (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\\\ 213749\(\text{HPV9-AS04-001}\) \(\text{WZA97329}\) \(\text{TFL Shells}\\\ \text{V3.0}\) \(\text{05FEB2024.docx}\)


Abbreviations: HPV = Human Papillomavirus. ECL = Electrochemiluminescence assay. PBNA = Pseudovirion-Based Neutralization Assay.

Deming regression model is fitted to the Anti-HPV IgG antibody concentration (ECL) with Anti-HPV Neutralizing titers (PBMA) as a covariate.

Deming's regression is computed by the log10-transformation of the antibody concentration and neutralizing titer. Samples testing below the LLOO or above ULOO in either assay were excluded from the analysis.

The dotted red line is the LLOQ value of xx.x for PBNA and xx.x for ECL.

The dashed red line is the ULOQ value of xx.x for PBNA and xx.x for ECL.

The solid line is based on the estimates obtained from Deming regression

#### Programming Notes

Timepoints will be Day 1 (blue circle), Month 2 (red plus), Month 3 (green cross) and Month 7 (black triangle).

Create each antigen and treatment group in separate plots

The dashed line is a reference plotted at 45 degrees

The x-axis is the PBNA value (Anti-HPV Neutralizing titers) while the Y axis will be the ECL value (Anti-HPV IgG antibody concentration.

Output ID: IM0009

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM


### Listing 16.2.1.1: Participants Disposition (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Listing 16.2.1.1 Participants Disposition Enrolled Set

| Participant<br>Identifier | Site<br>ID | Vaccine<br>Group | Date of<br>Vaccine<br>Dose | Completed /<br>Discontinued<br>the Study | Date of Completion / Discontinuation | Reason for Early<br>Discontinuation | Was Treatment<br>Unblinded by<br>Site? |
|---|---|---|---|---|---|---|---|
| Identifier xxxxxxxx | xx | Group HPV9 High HPV9 Medium HPV9 Low Gardasil 9 | Dose | the Study Completed Discontinued | / Discontinuation | AE requiring expedited reporting; AE no: xx Pregnancy Unsolicited AE; AE no: xx Withdrawal by participant; Specify: xxxxxxxx Migrated/moved from study area Lost to follow-up Study termination Subject discontinued | Yes: xxxxxxx |
| | | | | | | <pre>due to COVID-19 pandemic Other; Specify: xxxxx</pre> | |

Abbreviations: HPV = Human Papillomavirus. COVID-19 = Coronavirus disease 2019.

Programming Notes

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

Output ID: LS0001

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.1.2: Participants with Early Withdrawal or Discontinuation due to COVID-19 (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

# Listing 16.2.1.2 Participants with Early Withdrawal or Discontinuation due to COVID-19 Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site ID | Discontinue Treatment due to COVID-19 | Discontinue Study due to COVID-19 |
|---|---|---|---|
| | XX | Yes | Yes |
| XXXXXXX | XX | No | No |

Abbreviations: HPV = Human Papillomavirus. COVID-19 = Coronavirus disease 2019.

Programming Notes

Output ID: LS0002

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749\) (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\\\ 213749\(\text{HPV9-AS04-001}\) \(\text{WZA97329}\) \(\text{TFL Shells}\\\ \text{V3.0}\) \(\text{05FEB2024.docx}\)


### Listing 16.2.1.3: Participant Analysis Set (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.1.3
Participant Analysis Set
Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Date; Time of<br>Informed<br>Consent | Enrolled Set (ENR); If no, reason for exclusion | Exposed Set (ES); If no, reason for exclusion | Per Protocol Set (PPS); If no, reason for exclusion |
|---|---|---|---|---|---|
| xxxxxxx | xx | ddmmmyyyy;<br>hh:mm | Yes<br>No; xxxxxx | Yes<br>No; xxxxxx | Yes<br>No; xxxxxx |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0003

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749


### Listing 16.2.1.4: Inclusion and Exclusion Criteria at Enrolment (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant | | Inclusion/ Exclusion | |
|-------------|---------|----------------------|-----------------|
| Identifier | Site ID | Category Failed | Criteria Failed |
| XXXXXXX | XX | Inclusion | xxxxxxxxxxxxxx |
| | | Exclusion | |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0004

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749\) (HPV9)\Biostatistics\Documentation\SAP\Shells\\ GSK\\ 213749\) (HPV9-AS04-001)\(\quintiles\text{WZA97329\\ TFL\ Shells\\ V3.0\\ 05FEB2024.docx\)


### Listing 16.2.2.1: All Protocol Deviations (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.2.1 All Protocol Deviations Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Classification | Date of<br>Deviation | Deviation Category | Description | Exclusion<br>from Per<br>Protocol<br>Set? |
|---|---|---|---|---|---|---|
| xxxxxxx | XX | Important<br>Not important | ddmmmyyyy<br>ddmmmyyyy | Inclusion: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Xxxxxxxxxxxx | Yes<br>No |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0005

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.4.1: Demographics and Other Baseline Characteristics (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Listing 16.2.4.1 Demographics and Other Baseline Characteristics Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant | Site | Age | Year of | | | |
|---|---|---|---|---|---|---|
| Identifier | ID | (years) | Birth | Sex | Race | Ethnicity |
| xxxxxxx | XX | xx | УУУУ | Female | Black or African American | Hispanic of<br>Latino |
| | | XX | УУУУ | | American Indian or Alaska<br>Native | Not<br>Hispanic o<br>Latino |
| | | xx | УУУУ | | Asian<br>Native Hawaiian or other<br>Pacific Islander<br>White<br>Other | |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0006

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author: Version Date: 05FFB2024

### Listing 16.2.4.2: General Medical and Vaccination History (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

# Listing 16.2.4.2 General Medical and Vaccination History Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| | | | | System Organ Class; | |
|---|---|---|---|---|---|
| Participant<br>Identifier | Site ID | Diagnosis | Start /<br>End Date | Preferred Term; Description | Taking Medication Related to this Condition? |
| xxxxxxx | xx | xxxxxxxxx | ddmmmyyyy/<br>ddmmmyyyy | xxxxxxxxxxx<br>xxxxxxxxxxx<br>xxxxxxxxx | Yes |
| | | | ddmmmyyyy/<br>Ongoing | ***********<br>************************** | No |

Abbreviations: HPV = Human Papillomavirus. MedDRA = Medical dictionary for regulatory activities. MedDRA version xx.x.

Programming Notes

Output ID: LS0007

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.4.3: Prior and Concomitant Vaccinations (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

# Listing 16.2.4.3 Prior and Concomitant Vaccinations Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | ATC Classification; Preferred Term; Drug name (No.) | Indication | Prophy-<br>laxis | Dose | Unit | Frequency;<br>Route | Start (Onset<br>Day)/<br>End Date (End<br>Day) | Prior/<br>Concomitant? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | XX | xxxxxxxxxxx;<br>xxxxxxxxxxx;<br>xxxxxx (xx) | xxxxxxx | xxxxxx | xxxx | xxx | QID;<br>Oral | Ddmmmyyyy<br>(xx)/<br>ddmmmyyyy<br>(xx) | Concomitant |
| | | xxxxxxxxxxxx;<br>xxxxxxxxxxxx;<br>xxxxx (xx) | xxxxxxxx | xxxxxxx | XXXX | xxx | BID;<br>Topical | Ddmmmyyyy<br>(xx)/<br>Ongoing | Prior |
| | | xxxxxxxxxxxx;<br>xxxxxxxxxxx;<br>xxxxxx (xx) | | | | | TID;<br>xxx | | Concomitant |
| | | ,, | | | | | QD;<br>xxx | | |

Abbreviations: HPV = Human Papillomavirus. VV = Comparator vaccine. ATC = Anatomical therapeutic chemical. Prior vaccinations are vaccinations which started prior to the dose of study vaccination. Concomitant vaccinations are vaccinations which started on or after the day of the administration of study vaccination.

Programming Notes

Output ID: LS0008

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.4.4: Concomitant Medications (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

# Listing 16.2.4.4 Prior and Concomitant Medications Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | ATC Classification; Preferred Term; Drug name (No.) | Indication | Prophy-<br>laxis | Dose | Unit | Frequency;<br>Route | Start (Onset<br>Day)/<br>End Date (End<br>Day) | Prior/<br>Concomitant? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx | xxxxxxxxxxxx;<br>xxxxxxx (xx)<br>xxxxxxxxxxxxx;<br>xxxxxxxxxxxxx;<br>xxxxx (xx) +^<br>xxxxxxxxxxxxx;<br>xxxxxxxxxxxx;<br>xxxxxxxx | xxxxxxxx<br>xxxxxxxx | ***** | xxxx | xxx | QID;<br>Oral<br>BID;<br>Topical<br>TID;<br>xxx | Ddmmmyyyy (xx)/ ddmmmyyyy (xx) Ddmmmyyyy (xx)/ Ongoing | Concomitant Prior Concomitant |
| | | , | | | | | QD;<br>xxx | | |

Abbreviations: HPV = Human Papillomavirus. VV = Comparator vaccine. ATC = Anatomical therapeutic chemical.

 $^{\star}$  = Anti-pyretic medication, + = Antibiotic medications.  $^{\wedge}$  = Prophylactic medications.

Prior medications are medications which started prior to the dose of study vaccination.

Concomitant medications are medications which started on or after the day of the administration of study vaccination.

Programming Notes

Output ID: LS0009

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.5: Vaccine Administration (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.5 Vaccine Administration Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Vaccine Administered?<br>If no, reason | Date of Administration (Study Day) | Route;<br>Location | Kit<br>Number | Remain under observation? |
|---|---|---|---|---|---|---|
| xxxxxxx xx | XX | Yes | ddmmmyyyy (xx) | Intramuscular;<br>Arm Upper Left | xxxxx | Yes |
| | | No; Adverse Event (xx) No; not willing to be vaccinated No; Other: specify | | Intramuscular;<br>Arm Upper Right | | No |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0010

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


## Listing 16.2.6.1: Listing of anti-HPV IgG Antibody Concentration for each Participant (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### 

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant | | | anti-HPV Antibody | | |
|---|---|---|---|---|---|
| Identifier | Site ID | Visit | Concentration (mIU/mL) | Seropositive | Seroconversion |
| xxxxxxx | XX | Day 1 | xx | Yes | |
| | | Month 1 | | No | No |
| | | Month 2 | | | Yes |
| | | Month 3 | | | |
| | | Month 6 | | | |
| | | Month 7 | | | |
| | | Month 12 | | | |

Abbreviations: HPV = Human Papillomavirus.

Seropositive is defined as the appearance of antibodies (i.e, concentrations greater than or equal to xx = mIU/mL) in the serum of participants.

Seroconversion is defined as the appearance of antibodies (i.e, concentrations greater than or equal to xx = MU/mL) in the serum of participants seronegative before vaccination.

Programming Notes

Output ID: LS0011

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Author:


### Listing 16.2.6.2: Listing of anti-HPV IgG Neutralizing Antibody Titers for each Participant (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### Listing 16.2.6.2 Listing of anti-HPV IgG Neutralizing Antibody Titers for each Participant Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site ID | Visit | <pre>anti-HPV Antibody Titers (mIU/mL)</pre> | Seropositive | Seroconversion |
|---|---|---|---|---|---|
| | | | | - | |
| XXXXXXX | XX | Day 1 | XX | Yes | |
| | | Month 1 | | No | No |
| | | Month 2 | | | Yes |
| | | Month 3 | | | |
| | | Month 6 | | | |
| | | Month 7 | | | |
| | | Month 12 | | | |

Abbreviations: HPV = Human Papillomavirus.

Seropositive is defined as the appearance of antibodies (i.e, titer greater than or equal to xx mIU/mL) in the serum of participants.

Seroconversion is defined as the appearance of antibodies (i.e, titer greater than or equal to xx mIU/mL) in the serum of participants seronegative before vaccination.

Programming Notes

Output ID: LS0012

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.7.1: Solicited Administration Site Events (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

### Listing 16.2.7.1 Solicited Administration Site Events Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Date of<br>Assessment<br>(Study<br>Day) | Vaccine<br>dose | Injection<br>Site Pain?<br>If Yes,<br>severity | Injection Site Pain leading to Medical Attention | Redness at Injection Site? If Yes, size (mm), Grade | Redness leading<br>to Medical<br>Attention | Swelling at<br>Injection<br>Site? If<br>Yes, size<br>(mm), Grade | Swelling<br>leading to<br>Medical<br>Attention |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | XX | ddmmmyyyy<br>(Day x) | 1/2/3 | Yes; Mild/<br>Moderate/<br>Severe | None | Yes; xx,<br>Gx | None | Yes; xx, Gx | None |
| | | | | No | Hospitalization<br>ER Visit<br>Other | No | Hospitalization<br>ER Visit<br>Other | No | Hospitalization<br>ER Visit<br>Other |

Abbreviations: HPV = Human Papillomavirus. G1 = Mild, G2 = Moderate, G3 = Severe.

Programming Notes

Output ID: LS0013

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas | IOVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.7.2: Solicited Systemic Events (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.7.2 Solicited Systemic Events Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Date of<br>Assessment<br>(Study<br>Day) | Vaccine<br>dose | Highest<br>Daily<br>Temper-<br>ature,<br>Grade | Headache?<br>If Yes,<br>intensity | Myalgia?<br>If Yes,<br>Intensity | Arthralgia?<br>If Yes,<br>Intensity | Fatigue?<br>If Yes,<br>severity | Experience other serious symptoms? | Additional medications?; Additional vaccinations? | Day; Additi- onal Vaccin- ation; Date |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx | ddmmmyyyy<br>(Day x) | 1/2/3 | xx, Gx | Yes; Mild /<br>Moderate/<br>Severe | Yes; Mild /<br>Moderate /<br>Severe | Yes; Mild/<br>Moderate/<br>Severe | Yes;<br>Mild/<br>Moderate<br>/ Severe<br>No | Yes | Yes; Yes | Xx;<br>Xxxx<br>Xxxxx |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0014

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.7.3: Unsolicited Adverse Events (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.7.3
Unsolicited Adverse Events
Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | System Organ<br>Class;<br>Preferred Term;<br>AE term<br>(Vaccine Dose) | Start Date (Onset Day); End Date (Study Day) | Duration<br>(Days) | Severity;<br>Relationship<br>to Study<br>Treatment | Action Taken to Study Drug; Outcome | Potential<br>Immune-<br>Mediated<br>Disease<br>(pIMD)<br>event? | Serious;<br>If yes,<br>Criteria | Medical<br>Attention | COVID19? | Treatment<br>Given? If<br>Yes,<br>Treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx | xxxxxxxxx;<br>xxxxxxxxx;<br>xxxxxx (x) | ddmmmyyyy (x); ddmmmyyyy (x) | xx | Mild / Moderate/ Severe; Related / Not Related | xxxxx;<br>xxxxxxx | Yes | Yes; xxxx | Yes | Yes | No<br>Yes; xxxx |

Abbreviations: HPV = Human Papillomavirus. COVID19 = Coronavirus disease 2019. MedDRA = Medical dictionary for regulatory activities.

MedDRA version xx.x.

Unsolicited AEs include serious AEs.

Programming Notes

Output ID: LS0015

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

Document:


05FEB2024 Version Date:

### Listing 16.2.7.4: Unsolicited Adverse Events Leading to Withdrawal or Discontinuation from Study (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

#### 

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9 Potential Start Date System Organ (Onset Action Immune-Mediated Class; Day); End Taken to Severity; Treatment Preferred Term; Date Relationship Study Disease Serious; Given? If Participant Site (Study Duration to Study Drug; (DMIq) If yes, Medical AE term Yes, Identifier ID (Vaccine Dose) Day) (Days) Treatment Outcome event? Criteria Attention COVID19? Treatment Mild / ddmmmyyyy Yes No xxxxxx; Moderate/ (x); XXXXXXXX XXXXXXXXXX; Severe; XXXXXXX XX xxxxxxxxx; ddmmmyyyy XX Yes Yes; xxxx Yes Related / xxxxxx (x) (x) Not Related No No No Yes; xxxx

Abbreviations: HPV = Human Papillomavirus. COVID19 = Coronavirus disease 2019. MedDRA = Medical dictionary for regulatory activities.

MedDRA version xx.x.

Unsolicited AEs include serious AEs.

Programming Notes

Output ID: LS0016

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas| IOVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001) WZA97329 TFL Shells V3.0 05FEB2024.docx


### Listing 16.2.7.5: Serious Adverse Events (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.7.5 Serious Adverse Events Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| | | System Organ Class; | | |
|-------------|---------|------------------------|-----------|---|
| Participant | | Preferred Term; | | |
| Identifier | Site ID | AE Term (Vaccine Dose) | Country | |
| | | | | • |
| | | xxxxxxxxxxxxxxx; | | |
| | | xxxxxxxxxxxxxx; | | |
| XXXXXXX | XX | xxxxxxxxxxxxx (x) | XXXXXXXXX | |

Abbreviations: HPV = Human Papillomavirus. Serious AEs are expedited adverse events.

Programming Notes

Output ID: LS0017

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx

Version Number: 3.0 Author: Version Date: 05FFB2024

### Listing 16.2.7.6: All Serious Adverse Events Leading to Withdrawal or Discontinuation from Study (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant | | System Organ Class;<br>Preferred Term; | |
|-------------|---------|----------------------------------------|----------|
| Identifier | Site ID | AE Term (Vaccine Dose) | Country |
| | | xxxxxxxxxxxxxxx; | |
| | | xxxxxxxxxxxxxx; | |
| XXXXXXX | XX | xxxxxxxxxxxxx (x) | XXXXXXXX |

Abbreviations: HPV = Human Papillomavirus. Serious AEs are expedited adverse events.

Programming Notes

Output ID: LS0018

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.7.7: Potential Immune-Mediated Disease Events (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| | | System Organ Class; | |
|---|---|---|---|
| Participant | | Preferred Term; | |
| Identifier | Site ID | AE Term (Vaccine Dose) | Country |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| | | xxxxxxxxxxxxxxx; | |
| XXXXXXX | XX | xxxxxxxxxxxxx (x) | XXXXXXXXX |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0019

Author:

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9)\Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \(\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749\) (HPV9)\Biostatistics\Documentation\SAP\Shells\\
GSK\\\ 213749\(\text{HPV9-AS04-001}\) \(\text{WZA97329}\) \(\text{TFL Shells}\\\ \text{V3.0}\) \(\text{05FEB2024.docx}\)


### Listing 16.2.8.1: Laboratory Results (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.8.1 Laboratory Results Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Visit | Collection date | Lab test | Result | Unit | Reference<br>Range | Investigator<br>assessment | Grade |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx | Visit 1<br>Visit 2 | ddmmmyyyy | Leukocytes Erythrocyte Hemoglobin Platelets Neutrophils Lymphocytes Monocytes Eosinophils Basophils BUN AST ALT | xx | xx | Xx - xx<br>No | Normal Abnormal, not clinically significant Abnormal, clinically significant | Grade 1<br>Grade 2<br>Grade 3<br>Grade 4 |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0020

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas | IOVIA DDMMMYYYY HH:MM

\\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\ Document: GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.8.2: Pregnancies - Follow up Report (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.8.2

Pregnancies - Follow up Report
Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site<br>ID | Pregnancy outcome | Date of outcome | Method used for delivery | Number of neonates | Gestational weeks at birth / miscarriage / termination |
|---|---|---|---|---|---|---|
| xxxxxxx | xx | Live infant, no apparent congenital anomaly Live infant congenital anomaly Elective termination, no apparent congenital anomaly Elective termination congenital anomaly Spontaneous abortion, no apparent congenital anomaly Spontaneous abortion congenital anomaly Spontaneous abortion congenital anomaly Stillbirth, no apparent congenital anomaly Stillbirth congenital anomaly Ectopic pregnancy Molar pregnancy Lost to follow-up Pregnancy ongoing | ddmmmyyyy | Normal vaginal Caesarean section Forceps delivery Vacuum delivery | xx | xx |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### GlaxoSmithKline Biologicals SA PROTOCOL 213749 (HPV9)

Output ID: LS0021

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\quintiles.net\Enterprise\Apps\sasdata\SAS\SAS\GlaxoSmithKline\HPV\213749 (HPV9)\Biostatistics\Documentation\SAP\Shells\

GSK 213749(HPV9-AS04-001)\_WZA97329\_TFL Shells\_V3.0\_05FEB2024.docx


### Listing 16.2.8.3: Vital Signs (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.8.3 Vital Signs Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant<br>Identifier | Site ID | Visit | Assessment<br>date | Parameter (unit) | Result |
|---|---|---|---|---|---|
| Identifier | DICE ID | V1310 | date | rarameter (unit) | Nesure |
| xxxxxxx | xx | Day 1<br>Month 1<br>Month 2 | ddmmmyyyy | Systolic Blood Pressure (mmHg) Diastolic Blood Pressure (mmHg) Heart rate (bpm) | xx |
| | | Month 3<br>Month 6 | | Respiratory rate (breathes/min) | |
| | | Month 7 | | | |
| | | Month 12 | | | |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0022

[Source: \quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749


3.0

### Listing 16.2.8.4: Body Temperature (Enrolled Set)

GSK Vaccines Page X of Y

Study 213749 - DELIVERY DESIGNATION

Listing 16.2.8.4 Body Temperature Enrolled Set

Vaccine Group: HPV9 High / HPV9 Medium / HPV9 Low / Gardasil 9

| Participant | | | Assessment | | |
|---|---|---|---|---|---|
| Identifier | Site ID | Visit | date | Temperature (unit) | Route |
| xxxxxxx | XX | Day 1 | ddmmmyyyy | Xx C | Axilla |
| | | Month 2 | 1111 | Xx F | Oral cavity |
| | | Month 6 | | | Tympanic membrane |
| | | | | | Temporal artery |

Abbreviations: HPV = Human Papillomavirus.

Programming Notes

Output ID: LS0023

[Source: \\quintiles.net\Enterprise\Apps\sasdata\SASb\SAS\GlaxoSmithKline\HPV\213749

(HPV9) \Biostatistics\Filename.sas] IQVIA DDMMMYYYY HH:MM

PPD Version Number:

Author:

Version Nate: 05FEB2024

### **Certificate Of Completion** Envelope Id: PPD Status: Completed Subject: Complete with DocuSign: GSK\_213749(HPV9-AS04-001)\_WZA97329\_SAP\_Final\_v3.0\_02FEB2024.docx, GSK\_2... Project Code (Enter 0 for non-billable projects): WZA97329 IQVIA ID (Login ID): PPD **Business Unit: Global Business Operations** Source Envelope: Document Pages: 207 Signatures: 6 **Envelope Originator:** PPD Certificate Pages: 5 Initials: 0 AutoNav: Enabled Envelopeld Stamping: Disabled Time Zone: (UTC-08:00) Pacific Time (US & Canada) **Record Tracking** Holder: PPD Status: Original Location: DocuSign 2/5/2024 7:30:11 AM **Signature Signer Events Timestamp** PPD PPD Sent: 2/5/2024 7:34:34 AM Viewed: 2/8/2024 11:19:23 AM Security Level: Email, Account Authentication Signed: 2/8/2024 11:20:58 AM (Required) Signature Adoption: Pre-selected Style Signature ID: Using IP Address: PPD With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document I approve this document **Electronic Record and Signature Disclosure:** Not Offered via DocuSign PPD PPD Sent: 2/5/2024 7:34:34 AM Viewed: 2/5/2024 7:41:43 AM Signed: 2/5/2024 7:42:41 AM Security Level: Email, Account Authentication Signature Adoption: PPD (Required) Signature ID:

Using IP Address: PPD

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 11/13/2020 12:14:20 AM

ID: PPD

**Signer Events Signature Timestamp** PPD Sent: 2/5/2024 7:34:35 AM Viewed: 2/5/2024 11:24:02 AM Security Level: Email, Account Authentication Signed: 2/5/2024 11:26:38 AM (Required) Signature Adoption: Pre-selected Style Signature ID: PPD

Using IP Address: PPD

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document I approve this document

### Electronic Record and Signature Disclosure: Accepted: 7/24/2023 3:40:35 AM

ID: PPD

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 2/5/2024 7:34:35 AM |
| Certified Delivered Signing Complete Completed | Security Checked Security Checked Security Checked | 2/5/2024 11:24:02 AM<br>2/5/2024 11:26:38 AM<br>2/8/2024 11:20:58 AM |
| Signing Complete | Security Checked<br>Security Checked | 2/5/2024 11:24:02 AM<br>2/5/2024 11:26:38 AM |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents will be sent to you electronically**

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

### **How to contact IOVIA:**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

### 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

### 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.